

| CD NUMBER: F-15267 | VERSION: 2.0 | PAGE 1 of 2 |
|---|---|---|
| TITLE: Statistical Analysis Plan (SAP)/Initiat | ion of Programming/SA | AP Addendum |

TITLE: Statistical Analysis Plan (SAP)/Initiation of Programming/SAP Addendum

Type of Approval (select one):  $\square$  SAP  $\square$  Initiation of Programming SAP

☐ SAP Addendum

| <b>Sponsor Name:</b> | Immutep S.A.S. | | |
|---|---|---|---|
| Sponsor<br>Protocol/<br>CIP ID: | TACTI-002<br>(IMP321-P015);<br>Keynote-PN798 | Fortrea Study<br>ID: | 41887 |
| SAP text filename: | TACTI-002_(P015)_Version_3_Final_SAP_31Jan2024 | | |
| TFL shells filename: | TACTI-002_(P015)_Version_3_Final_SAP_Shells_31Jan2024 | | |
| Version: | Version 3 | Date: | 31JAN2024 |

## Fortrea Approval(s):

**Lead Statistician** 

| Approval Signature Print Name Date | PPD |
|------------------------------------|-----|
| Not applicable | |
| _ | |

## **Sponsor Approval(s):**

By signing below when the statistical analysis plan (SAP) is considered final, the signatories agree to the analyses to be performed for this study and to the format of the associated tables, figures, and listings (TFLs). Once the SAP has been signed, programming of the Analysis Dataset Model (ADaM) datasets and TFLs based on these documents can proceed. Any modifications to the SAP text and TFL shells made after signing may result in a work-scope change.



TITLE: Statistical Analysis Plan (SAP)/Initiation of Programming/SAP Addendum
Approval Form



Approval
Signature
Print Name
Date



## Immutep S.A.S.

## STATISTICAL ANALYSIS PLAN

Protocol: TACTI-002 (IMP321-P015); Keynote-PN798

EUDRACT: 2018-001994-25

**Treatment:** eftilagimod alpha (efti, eftilagimod alfa, IMP321, LAG3-Ig)

pembrolizumab (Keytruda®; MK-3475)

TACTI-002 (Two ACTive Immunotherapeutics): A multicenter, open label, Phase II study in patients with previously untreated unresectable or metastatic non-small cell lung cancer (NSCLC), or recurrent PD-X refractory NSCLC or with recurrent or metastatic squamous head and neck cancer (HNSCC) receiving the soluble LAG-3 fusion protein eftilagimod alpha (IMP321) in combination with pembrolizumab (PD-1 antagonist)

| Author: | PPD |
|------------------|----------------------------------|
| Document Status: | Version 3 |
| Version Dates: | Version 1 Draft 1: 31JAN2020 |
| | Version 1 Draft 2: 01JUL2020 |
| | Version 1 Draft 3: 23OCT2020 |
| | Version 1 Final Draft: 29OCT2020 |
| | Version 1 Final: 29OCT2020 |
| | Version 2 Final: 05SEP2022 |
| | Version 3 Draft 1: 27OCT2023 |
| | Version 3 Draft 2: 13DEC2023 |
| | Version 3 Draft 3: 03JAN2024 |
| | Version 3 Final: 31JAN2024 |
| Pages: | 77 |

#### STATEMENT OF CONFIDENTIALITY

The information contained herein is expressly subject to the terms and conditions of the Confidentiality Agreement by and between Chiltern and Immutep.

TPBS001 Version 6 (based on TPQA036 Version 2)


Effective Date: 15<sup>th</sup> March 2017 Prior Effective Date: 9<sup>th</sup> October 2016

SAP Version 3, Final  31Jan2024



# **Contents**

| A | BBREVIATION | <b>NS</b> | ••••• | 5 |
|---|---|---|---|---|
| 1 | INTRODUC | TION | ••••• | 8 |
| 2 | STUDY OBJ | JECTIVES | ••••• | 9 |
| | | | | 9 |
| | | | | 9 |
| | | | | 10 |
| 3 | | | | 11 |
| 3 | | | | |
| | | | | 11 |
| | | | | 12 |
| | | | | 14 |
| | • | • | | |
| | • | | | 16 |
| | | | | 16 |
| | | | | of Cycles 1, 5 and 916 |
| | 3.3.7 Subje | cts Participating in PK I | Part Only - Days | 2, 3 4 and 5 of Cycles 1, 5 and 9 |
| | - ' | 19 to 35 Day 1 (Every 3 | Weeks) | 17 |
| | | • | | |
| | | _ | | 18 |
| | | <u> </u> | | |
| | | | | 19 |
| | | | | 20 |
| | | | | 20 |
| | | | | 20 |
| | | • | | 21 |
| | | - | | 21 |
| | <i>J V</i> | _ | | 21 |
| | 3.7 RANDOM | MIZATION | | 22 |
| | 3.8 BLINDIN | G | | 22 |
| | 3.9 SAMPLE | Size | | 22 |
| 4 | STATISTIC | AL METHODOLOGY | | 23 |
| • | | | | 23 |
| | | | | 24 |
| | | | | 24 |
| | | | | 25 |
| | | | | 27 |
| | | | | 28 |
| | PBS001 Version 6<br>pased on TPQA036 \ | | ONFIDENTIAL | Effective Date: 15 <sup>th</sup> March 2017<br>Prior Effective Date: 9 <sup>th</sup> October 2016 |
| ν, | acca on it water | 3.31311 <i>L</i> ) | | Endouve Date. 5 October 2010 |



TACTI-002 (IMP321-Sponsor: Immutep S.A.S. **Protocol Number:** P015); Keynote-PN798 4.8 4.9 Primary Efficacy Endpoint: iORR according to iRECIST ......30 4.9.2.1 4.9.2.2 Secondary Efficacy Endpoint: Disease Control Rate (DCR) According to Secondary Efficacy Endpoint: Progression Free Survival (PFS) According 4.9.2.3 Secondary Efficacy Endpoint: Duration of Response (DoR) according to 4.9.2.4 Secondary Efficacy Endpoint: Time to Response (TTR) According to 4.9.2.5 4.9.2.6 4.9.3 Exploratory Efficacy Endpoint Analyzes .......36 Exploratory Efficacy Endpoint: Circulating biomarkers.......36 4.9.3.1 4.9.3.2 4.9.3.3 Other Exploratory Endpoints ......37 4.9.4 4.9.4.1 4.9.4.2 4.10 4.11 4.11.1 4.11.2 Overall Survival (OS) by Response (Investigator assessment only)........41 TUMOR GROWTH KINETICS .......41 4.12 4.13 SAFETY ANALYSIS .......42 4.13.1 Adverse Events 43 4.13.2 4.13.3 Vital Signs 50 4.13.4 ECG Results 50 4.13.5 4.13.6 4.14 Center Effects 51 4.14.1 4.15 4.16 4.17 4.18 4.18.1 4.18.2 4.18.3 ALGORITHMS/SAS CODES 54 TABLES AND LISTINGS ......56 5.1 TPBS001 Version 6 CONFIDENTIAL Effective Date: 15th March 2017 (based on TPQA036 Version 2) Prior Effective Date: 9th October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
| 5.2 C | ONVENTIONS | | 56 |
| | | | 57 |
| 5.4 L | STINGS | | 65 |
| 5.5 F | GURES | | 67 |
| 5.6 A | PPENDICES | | 71 |
| <i>5.6.1</i> | Tumor growth kinetics anal | lysis in Part B - List of | patients and their lesions .71 |
| <i>5.6.2</i> | Subgroup for Part B (Prior | Therapy anti-PD-(L)1- | - <b>based – cat)</b> 76 |
| 5.7 R | EFERENCES | | 77 |



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

# **Abbreviations**

| AE | Adverse Event |
|---|---|
| ALC | |
| | Absolute Lymphocyte Count |
| ALT | Alanine Aminotransferase |
| ALK | Anaplastic Lymphoma Kinase |
| AR | All Randomized |
| AST | Aspartate Aminotransferase |
| BICR | Blinded Independent Central Reviewer |
| BMI | Body Mass Index |
| BOR | Best Overall response |
| BP | Blood Pressure |
| CPS | Combined positivity score |
| CR | Complete Response |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CXCL-10 | C-X-C motif chemokine 10 |
| DBP | Diastolic Blood Pressure |
| DCR | Disease Control Rate |
| DIAG | Data Monitoring Committee |
| DMC | Data Monitoring Committee |
| DMC | Duration of Response |
| DOR | Duration of Response |
| DOR<br>EAS | Duration of Response Evaluable Analysis Set |
| DOR<br>EAS<br>ECG | Duration of Response Evaluable Analysis Set Electrocardiogram |
| DOR EAS ECG ECI | Duration of Response Evaluable Analysis Set Electrocardiogram Events of clinical interest |
| DOR EAS ECG ECI ECOG | Duration of Response Evaluable Analysis Set Electrocardiogram Events of clinical interest Eastern Cooperative Oncology Group |
| DOR EAS ECG ECI ECOG eCRF | Duration of Response Evaluable Analysis Set Electrocardiogram Events of clinical interest Eastern Cooperative Oncology Group Electronic Case Report Form |
| DOR EAS ECG ECI ECOG eCRF EGFR | Duration of Response Evaluable Analysis Set Electrocardiogram Events of clinical interest Eastern Cooperative Oncology Group Electronic Case Report Form Epidermal Growth Factor Receptor |
| DOR EAS ECG ECI ECOG eCRF EGFR EOC | Duration of Response Evaluable Analysis Set Electrocardiogram Events of clinical interest Eastern Cooperative Oncology Group Electronic Case Report Form Epidermal Growth Factor Receptor End of Combination |
| DOR EAS ECG ECI ECOG eCRF EGFR EOC | Duration of Response Evaluable Analysis Set Electrocardiogram Events of clinical interest Eastern Cooperative Oncology Group Electronic Case Report Form Epidermal Growth Factor Receptor End of Combination End of Treatment |
| DOR EAS ECG ECI ECOG eCRF EGFR EOC | Duration of Response Evaluable Analysis Set Electrocardiogram Events of clinical interest Eastern Cooperative Oncology Group Electronic Case Report Form Epidermal Growth Factor Receptor End of Combination |




| HIV | Human Immunodeficiency virus |
|-----------|----------------------------------------------|
| HNSCC | Head and neck squamous cell carcinoma |
| HPV | Human papilloma virus |
| Hr | Hour |
| ICF | Informed Consent Form |
| i control | Reference to iRECIST guideline |
| iCPD | Confirmed progressive disease |
| IEC | Independent Ethics Committees |
| IFN-γ | Interferon gamma |
| IMP | Investigational Medicinal Product |
| irAEs | Immune-Related Adverse Events |
| IRB | Institutional Review Boards |
| iUPD | Unconfirmed progressive disease |
| kg | Kilogram |
| L | Liter |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| Min | Minimum |
| mL | milliliter |
| NCI | National Cancer Institute |
| NSCLC | Non-small cell lung cancer |
| ORR | Overall response rate |
| OS | Overall survival |
| PD | Progressive disease |
| PD-L1 | Programmed cell death ligand 1 |
| PFS | Progression free survival |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PR | Partial Response |
| RBC | Red Blood Corpuscle |




| Sponsor: Immutep S.A.S. Protocol Number: TACTI-002 (IMP321-P015); Keynote-PN798 | Immutep S.A.S. Protocol Number: TACTI-002 (IMP321 P015); Keynote-PN7 |
|---|---|
|---|---|

| RECIST | Response evaluation criteria in solid tumors |
|--------|----------------------------------------------|
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SD | Stable Disease |
| SMQ | Standardized MedDRA Queries |
| TPR | Timepoint to Response |
| TPS | Tumor proportion score |
| TTR | Time to response |
| WBC | White blood cell |




## 1 Introduction

This document presents the statistical analysis plan (SAP) for Immutep, Protocol No. TACTI-002 (IMP321-P015); Keynote-PN798: TACTI-002 (Two ACTive Immunotherapeutics): A multicenter, open label, Phase II study in patients with previously untreated unresectable or metastatic non-small cell lung cancer (NSCLC), or recurrent PD-X refractory NSCLC or with recurrent or metastatic squamous head and neck cancer (HNSCC) receiving the soluble LAG-3 fusion protein eftilagimod alfa (IMP321) in combination with pembrolizumab (PD-1 antagonist).

Version 1 of this analysis plan is based on the final protocol version 3.0 dated 28<sup>th</sup> July 2020 and electronic case report form (eCRF) version 5 dated 6<sup>th</sup> June 2019.

Version 2 of this analysis plan is based on the final protocol version 4.0 dated 30<sup>th</sup> April 2021 and electronic case report form (eCRF) version 6 dated 23<sup>rd</sup> March 2021.

Version 3 of this analysis plan is based on the final protocol version 5.0 dated 18<sup>th</sup> Aug 2023 and electronic case report form (eCRF) version 6 dated 23<sup>rd</sup> March 2021. This version is also updated to include additional analyzes and subgroup variables. Certain analyzes presented in Version 2 have been deleted in the list of outputs in section 5.

The SAP provides the description of every analysis including interim, primary and follow up analyzes.




| Sponsor: | Immutep S.A.S. | i Protocol illimper. | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

2 Study Objectives

The primary objective of this study is:

• To evaluate the response rate of eftilagimod alfa in combination with pembrolizumab in subjects with advanced, metastatic, recurrent NSCLC and HNSCC.

The secondary objectives of this study are:

- To evaluate the safety and tolerability of eftilagimod alfa when combined with pembrolizumab.
- To further evaluate the antitumor activity of eftilagimod alfa when combined with pembrolizumab.
- To assess the pharmacokinetic and immunogenic properties of eftilagimod alfa.

The exploratory objective of this study is:

- To identify and characterize relevant biomarkers.
- To further characterize the antitumor activity of eftilagimod alfa in combination with pembrolizumab.

## 2.1 Primary Endpoints

The primary endpoint of this study is:

• To determine best overall response rate (ORR) according to iRECIST.

## 2.2 Secondary Endpoints

The secondary endpoints of this study are:

- Safety profile in terms of frequency, severity and duration of adverse events (AEs), serious adverse events (SAEs) according to the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V5.0, events of clinical interest (ECI) and abnormalities in vital signs, physical examination, 12-lead electrocardiogram (ECG) and safety laboratory assessments.
- To assess time to response (TTR) and duration of response (DOR) according to iRECIST and RECIST 1.1.
- To assess ORR according to RECIST 1.1.
- To assess the disease control rate (DCR) according to iRECIST and RECIST 1.1.
- To assess progression free survival (PFS) and overall survival (OS).
- To assess occurrence and nature of anti- eftilagimod alfa-specific antibodies.
- To assess the plasma concentration time profile and derived PK parameters which may include but will be not limited to area under the curve (AUC), peak plasma concentration (Cmax), time to reach Cmax (tmax), systemic clearance (CL), elimination half-life (t1/2) and volume of distribution (VD) of eftilagimod alfa.



## 2.3 Exploratory Endpoints

The exploratory endpoints of this study are:

- To assess programmed cell death ligand 1 (PD-L1) expression assessed by central laboratory.
- CC
- To assess Gene signature according to PanCancer Immune code set assessed by a central laboratory.
- To assess circulating level of Helper T Cells Type 1 (Th1) biomarkers [i.e., interferon gamma (IFN- $\gamma$ ), C-X-C motif chemokine 10 (CXCL-10)] assessed by a central laboratory.
- · CCI




# 3 Study Design

## 3.1 Discussion of Study Design

The study was designed according to Simon's optimal two-stage design<sup>[1]</sup>. During the first stage of the study the number of N1 subjects were recruited for each indication into this multicenter, open label, phase II study. In case there were more responses than threshold r1 observed in subjects recruited in the initial stage (N1), additional subjects (N2) were to be recruited. Following the completion of the initial stage, the decision to recruit the additional subjects (N2) was taken by the Data Monitoring Committee (DMC), as described later.

| Indication | Threshold r1 | Initial No of pts<br>(N1) | Add. No. of pts (N2) | N total |
|---|---|---|---|---|
| NSCLC 1 <sup>st</sup> line | 4 | 17 | 19 | 36 |
| NSCLC 2 <sup>nd</sup> line | 1 | 23 | 13 | 36 |
| HNSCC | 2 | 18 | 19 | 37 |

In case ORR in any part met a predefined threshold, an extension of this cohort could be set up to combine the patients of stages 1, 2, and newly enrolled patients to provide a reasonable basis in sample size considerations for further clinical studies. For sample size considerations in the extension phase, please refer to the section "sample size calculations" in the synopsis and Chapter 10 of the protocol.

To be eligible for participation, subjects must have had either:

<u>Part A:</u> Histologically- or cytologically-confirmed diagnosis of NSCLC stage IIIB not amenable to curative treatment (unresectable) or stage IV not amenable to Epidermal Growth Factor Receptor (EGFR)/ Anaplastic Lymphoma Kinase (ALK) based therapy, treatment naïve for advanced/metastatic disease.

Note: subjects who received durvalumab or any other PD-1 or PD-L1 therapy as maintenance therapy to the adjuvant chemotherapy regimen and hence are not naïve to anti-PD-X agents, could be recruited provided that all other necessary requirements were met.

<u>Part B:</u> histologically- or cytologically-confirmed diagnosis of NSCLC after failure of first-line treatment (for metastatic/advanced disease) with at least 2 cycles of any PD-1/PD-L1 therapy (e.g., nivolumab, pembrolizumab, avelumab, durvulumab, etc.) alone, or in combination with any other immunotherapeutic or chemotherapy given as part of first-line treatment.

Note: Failure on therapy is defined as progress acc. to RECIST 1.1 and would require confirmation by a second assessment no less than four weeks from the first documented PD in the absence of rapid clinical progression. If patients discontinued PD-1/PD-L1 after being treated for at least 2 cycles for reasons other than progression, they could enroll in the study if initial progression occurred within 12 weeks after end of PD-1/PD-L1 therapy and progression was confirmed. Only patients receiving treatment in true second-line setting could be enrolled to Part B. Patients who received durvalumab or any other PD-1 or PD-L1 therapy as part of their adjuvant therapy and no other PD-1/PD-L1 therapy in the first line treatment were not eligible for Part B.


Effective Date: 15th March 2017

Prior Effective Date: 9th October 2016



| Sponsor: | Immutep S.A.S. | I Protocol Killmaner. | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Note: In Parts A and B subjects with neuroendocrine or sarcomatoid NSCLC tumor types were not eligible. Patients with undifferentiated lung carcinoma with certain neuroendocrine features could be recruited.

<u>Part C:</u> Histologically- or cytologically-confirmed recurrent disease not amenable to curative treatment with local or systemic therapy, or metastatic (disseminated) HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx that was considered incurable by local therapies after failure of prior platinum-based therapy.

Note: in all three parts subjects would be enrolled regardless of their PD-L1 expression.

## 3.2 Study Treatment

### Part A+B+C:

Subjects received pembrolizumab and effilagimod alfa starting from cycle 1 day 1 as follows:

- 200 mg pembrolizumab every 3 weeks intravenously (IV) (30 min) for up to 35 cycles; 1 cycle = 3 weeks;
- 30 mg of eftilagimod alfa (efti, IMP321) every 2 weeks subcutaneously (s.c.) for the first six months (until including cycle 8) and shifted to every three weeks s.c. thereafter (cycle 9 to 18); 1 cycle = 3 weeks.



Legend: 1 cycle = 3 weeks; q2w = every 2 weeks; q3w = every 3 weeks.

Figure 1: Study flow chart for Part A, B and C.

Screening of subjects for eligibility to enter this study was done in the three weeks prior to cycle 1 day 1. Subjects were enrolled in parallel except for the first three subjects in each part who were enrolled at least 1 week apart. A subject stayed on treatment until disease progression, unacceptable toxicity, completion of 35 cycles of pembrolizumab (~2 yrs.; completion of study treatment) or discontinuation for any other reason. Three (3) weeks after end of the combination therapy (cycle 18) end of combination (EOC) therapy assessments were to be performed. Three (3) weeks after end of any study treatment (cycle 35) an end of treatment (EOT) visit was to be performed. Upon start of study treatment, subjects will be followed for PFS and OS. PFS will be radiologically assessed at the study sites until PD, death, withdrawal of consent, loss to follow-up, or until the end of the study, whichever occurs first.

Radiological assessment will be performed at intervals of 9 weeks until week 36 (week 9, 18, 27, 36) and every 12 weeks thereafter (after week 36). OS will be monitored until death, withdrawal of consent, loss to follow-up or until the end of the study, whichever occurs first.



| Sponsor: | Immutep S.A.S. | I Protocol Killmaner. | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Measurability will be assessed according to iRECIST. Response to treatment and treatment decisions will be assessed according to iRECIST. Objective response [partial response (iPR), complete response (iCR)] should be confirmed by a repeat imaging assessment at least 4 weeks after the first response is observed. Per iRECIST, disease progression should be confirmed 4 to 8 weeks after site-assessed first radiologic evidence of unconfirmed progressive disease (iUPD). Subjects who have iUPD should stay on treatment (if clinically stable) until progression is confirmed (confirmed progressive disease (iCPD), provided they have met the conditions detailed in protocol Section 8.1.3.

Radiological scans and related information will be evaluated at the study sites for treatment decision and for primary objective but will be collected for potential later central evaluation by blinded independent radiologists.

Safety procedures are described in Section 9 of the protocol.

The study agents must be administered in a clinical setting where emergency resuscitative equipment and personnel trained in the management of anaphylaxis are immediately available to treat systemic reactions under the direct supervision of the physician.

The DMC reviewed available safety data of all subjects (part A-C) after 18 subjects completed at least two cycles (6 weeks) of therapy. In addition, the DMC reviewed the efficacy and safety data after the last subject N1 was enrolled or the minimum number of responses is reached for each part of the study, whatever was first. Subjects included in this decision needed at least one tumor imaging after treatment was initiated. The DMC gave a recommendation for each part of the study whether stage 2 could be opened. The details are described in the DMC charter.

Furthermore, the DMC will monitor safety and efficacy data at regular intervals and in accordance with the DMC charter. The DMC may recommend stopping/changing the study if at any time during the trial there are unacceptable adverse events or safety concerns. Unless immediate action is required to protect the safety and well-being of study subjects, the sponsor will consult with appropriate regulatory authorities prior to early termination of the study based on any DMC recommendation.

The Sponsor could, after careful evaluation, decide to temporarily suspend or prematurely discontinue this study either at a single site, multiple sites or at all sites at any time for reasons including but not limited to, incidence or severity of AEs in this study that indicate a potential health hazard to study subjects, unacceptable safety concerns, unfavorable risk/benefit ratio, ethical issues, inaccurate or incomplete data recording, noncompliance or unsatisfactory enrolment with respect to quality or quantity and decision by the Sponsor to suspend or discontinue testing, evaluation, or development of the product.

Subject safety will be monitored at study level (within the DMC) and on substance level (Immutep safety monitoring board). The recommendation of the above committees will be taken into consideration in such decisions of the Sponsor. The Investigators will be notified by the sponsor if the study is terminated or placed on hold. The relevant Independent Ethics Committees (IEC) / Institutional Review Boards (IRB) and health authorities will also be informed according to applicable regulatory requirements.

The end of study is defined 36 months after last patient first visit.




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

3.3 Study Schedule

Subjects were screened for suitability for participation in the study within -21 to -1 days prior to the first administration of pembrolizumab and effilagimod alfa (Visit 1: Day 1 of Cycle 1).

Screening assessments will include:

- Obtaining written informed consent prior to any study specific procedure (including screening procedures) being performed. Note: Subject can be consented up to 35 days before cycle 1 day 1 to allow planning of fresh tumor biopsy and/or perform computed tomography (CT) scan for assessment of eligibility at screening (the latter for Part B only). All screening assessments including the biopsy or confirmatory tumor assessment for Part B (to confirm progression) itself are still to be performed between -21 days and -1.
- Check for every inclusion and exclusion criteria.

Re-screening in the case of isolated out-of-range lab results during the screening period may be allowed on a case-by-case basis. The investigator must receive the approval from the Medical Monitor for each case beforehand.

Each treatment cycle consisted of 3 weeks. After enrolment, each subject was to visit the hospital according to the schedule of assessments.

### 3.3.1 Screening (Day: -21 to -1)

- Confirmation of written informed consent form (ICF) of subject and Investigator (including ICF for PK sampling where applicable);
- Inclusion & exclusion criteria;
- Medical history & demographics;
- Physical examination including height and weight;
- Eastern Cooperative Oncology Group (ECOG) performance status;
- AEs:
- Prior Concomitant medications/procedures;
- 12- lead ECG (single);
- Vital signs;
- Laboratory testing
  - Hematology, biochemistry, coagulation and urinalysis;
  - Thyroid function test;
  - o Pregnancy;
  - Human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis
     C virus (HCV) (where applicable);
  - o Gene expression profiling.
- Radiological assessment;



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

• Tumor tissue sample.

## 3.3.2 Day 1 of Cycles 1 to 8

Prior to pembrolizumab and eftilagimod alfa (efti, IMP321) administration:

- Confirmation of eligibility and assignment to treatment ONLY cycle 1;
- Physical examination including weight;
- ECOG performance status;
- AEs;
- Concomitant medication/procedures;
- 12-lead ECG;
- Vital signs;
- Laboratory testing:
  - hematology, biochemistry, coagulation and urinalysis;
  - o Thyroid function tests ONLY Cycle 2, 4, 6 and 8;
  - Autoantibodies ONLY pre-dose cycle 1;
  - o Pregnancy testing (urine);
  - Anti-drug (efti) antibodies ONLY pre-dose cycle 1 and 5;
  - o Th1 biomarker ONLY pre-dose Cycle 1 and 5;
  - o Gene expression profile ONLY pre-dose Cycle 5.
- Pembrolizumab infusion;
- For subjects who participate in the PK sampling please see Sections 3.3.6 and 3.3.7;
- Efti injection  $\geq$  30 minutes after pembrolizumab infusion was completed ONLY cycle 1, 3, 5 and 7.

Subjects should remain in the ward for a minimum of 30 min after last study drug administration.

## 3.3.3 Day 8 of Cycles 2, 4, 6 and 8

Prior to eftilagimod alfa (efti, IMP321) administration:

- AEs;
- Concomitant medication/procedures;
- Vital signs;
- Laboratory testing:
  - o Anti-drug (efti) antibodies ONLY pre-dose Cycle 2.
- Efti administration.

Subjects should remain in the ward for a minimum of 30 min after injection.




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

## 3.3.4 Day 15 of Cycles 1, 3, 5 and 7

Prior to eftilagimod alfa (efti, IMP321) administration:

- AEs;
- Concomitant Medication/procedures;
- Vital signs;
- Laboratory testing:
  - o Anti-drug (efti) antibodies ONLY pre-dose Cycle 3.
- Efti administration.

Subjects should remain in the ward for a minimum of 30 min after injection.

## 3.3.5 Day 1 of Cycles 9 to 18

Prior to pembrolizumab and eftilagimod alfa (efti, IMP321) administration:

- Physical examination including weight;
- ECOG performance status;
- AEs;
- Concomitant medication/procedures;
- 12-lead ECG;
- Vital signs;
- Laboratory tests:
  - o Hematology, biochemistry, coagulation and urinalysis;
  - o Thyroid function test ONLY cycle 10, 12, 14, 16 and 18;
  - o Pregnancy testing (urine);
  - Autoantibodies ONLY Cycle 9;
  - o Anti-drug (efti) antibodies ONLY pre-dose Cycle 9 and 13;
  - o Th1 biomarkers ONLY Cycle 9 and 13.
- Pembrolizumab infusion.
- For subjects who participate in the PK sampling please see Sections 3.3.6 and 3.3.7.
- Efti injection ≥30 minutes after pembrolizumab infusion was completed.

Subjects should remain in the ward for a minimum of 30 min after last study drug administration.

### 3.3.6 Subjects Participating in PK Part Only - Day 1 of Cycles 1, 5 and 9

Prior to effilagimod alfa (effi, IMP321) administration: blood sampling pre-dose.

After administration: blood sampling at 1, 2, 4 and 8h post-injection.




## 3.3.7 Subjects Participating in PK Part Only - Days 2, 3 4 and 5 of Cycles 1, 5 and 9

After administration: blood sampling at 24, 48, 72, 96 hours post-injection.

Adverse events and concomitant medications are to be recorded as well.

## 3.3.8 Cycle 19 to 35 Day 1 (Every 3 Weeks)

Prior to pembrolizumab administration:

- Physical examination including weight;
- ECOG performance status;
- AEs;
- Concomitant medication/procedures;
- 12-lead ECG;
- Vital signs;
- Laboratory tests:
  - o Hematology, biochemistry, coagulation and urinalysis;
  - Pregnancy testing (urine);
  - o Thyroid function test ONLY cycle 20, 22, 24, 26, 28, 30, 32 and 34;
  - Autoantibodies ONLY Cycle 19;
  - o Anti-drug (efti) antibodies ONLY Cycle 19;
  - o Th1 biomarkers ONLY Cycle 19.
- Pembrolizumab infusion.

#### 3.3.9 End of Treatment Visit

All subjects are scheduled to receive 8 cycles of combined pembrolizumab every 3 weeks and efti every 2 weeks followed by a further 10 cycles of pembrolizumab and efti every 3 weeks. Thereafter pembrolizumab will be given every 3 weeks (cycle 19 till cycle 35) unless of the previously specified reasons occur. An EOT visit will be performed 3 weeks ( $\pm$  7 days) after the last dose of any study treatment. The subjects should then continue with PFS follow-up or OS follow-up dependent on the status of their disease.

The following assessments will be performed at the EOT visit:

- AEs;
- Concomitant medication/procedures;
- Physical examination including weight;
- ECOG performance status;
- 12-lead ECG;
- Vital signs;

SAP Version 3, Final

• Laboratory tests:


Effective Date: 15th March 2017

31Jan2024



| Sponsor: Immutep S.A. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|
|---|---|---|

Hematology, biochemistry, coagulation and urinalysis;

- o Pregnancy testing (urine);
- Thyroid function test;
- Autoantibodies;
- Anti-drug (efti) antibodies (ADA);
- o Th1 biomarkers.

#### 3.3.10 PFS - Follow-Up

Subjects who complete all study Treatment Visits without documented PD will attend PFS Follow-Up Visits every 12 weeks (± 9 days) until PD, start of next anti-cancer therapy, pregnancy, withdrawal of consent, loss to follow-up, death from any cause, or the end of the study (whichever occurs first).

For subjects who prematurely discontinue treatment for any reason except PD and do not receive any other anti-cancer therapy or any other investigational therapy, PFS Follow-Up Visits will occur every 9 weeks until week 36 after treatment assignment (the start of the treatment, Cycle 1 Day1) and every 12 weeks after week 36 dependent on the most recent radiological assessment prior to discontinuation.

At each PFS Follow-Up Visit, the following will be performed:

- Radiological assessment;
- ECOG performance status and body weight;
- AE follow-up.

Note: Once a subject starts new line of anti-cancer therapy, the subject will be followed up for OS. Details on the next anti-cancer therapies will be recorded.

#### **3.3.11 OS - Follow-Up**

After documented PD, or after start of any next line of anti-cancer therapy, the subject will be followed up for survival every 12 weeks ( $\pm$  4 weeks) until end of study, lost to follow-up, withdrawal of consent or death whatever occurs first. The first overall survival visit will take place 12 weeks after the last visit of the treatment phase (EOC, EOT) or PFS follow up whatever was last. The visit can be performed via a telephone call. If necessary, subjects may be contacted occasionally outside of this follow up (FU) window.

Subjects who progress while on study treatment may receive any other next line of therapy, as clinically indicated, after performing the EOT visit. Subject who do not progress and complete the study treatment period (i.e., reach the end of cycle 35 without progression) may receive any other next line of therapy, as clinically indicated, after performing the EOT visit. In both cases this is to be recorded during overall survival follow-up. Additionally, any details on the next anti-cancer therapies and their duration/outcome will be recorded.

#### 3.3.12 Unscheduled Visits

Additional unscheduled visits may be conducted to assess adverse events or to evaluate disease status or for any other reason according to the Investigator's clinical judgment. These visits will be documented in the eCRF.




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

#### 3.4 Concomitant Medication

Medications or vaccinations specifically prohibited in the exclusion criteria (including the timeframe mentioned there) are not allowed during the ongoing trial. If there is a clinical indication for any medication or vaccination specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The investigator should discuss any questions regarding this with the Medical Monitor. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician. However, the decision to continue the subject on study treatment requires the mutual agreement of the investigator, the Sponsor and the subject.

Listed below are specific restrictions for concomitant therapy or vaccination during the course of the study:

- Antineoplastic systemic chemotherapy or biological therapy;
- Immunotherapy not specified in this protocol;
- Chemotherapy not specified in this protocol;
- Investigational agents other than pembrolizumab and/or efti;
- Radiation therapy;

Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be allowed at the investigator's discretion.

- Live vaccines within 30 days prior to the first dose of study treatment, while participating in the study and four months after the last dose of Investigational Medicinal Product (IMP). Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed;
- Systemic glucocorticoids for any purpose other than (1) to modulate symptoms from an AE that is suspected to have an immunologic etiology or (2) to treat an AE of not immunologic etiology, only for a short course (i.e. no longer than 10 days) and if that is in line with the site's SOC. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalents are permitted in the absence of active auto-immune disease. In case of doubt, the study Medical Monitor should be contacted.

Subjects who, in the assessment of the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the study treatment.

All treatments that the Investigator considers necessary for a subject's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care.

Acceptable concomitant therapy is defined as follows:



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

• Subjects may receive supportive care including but not limited to antibiotics, analgesics, transfusion of blood products, anti-diarrheal medication or laxatives according to local clinical practice and the approved pembrolizumab label.

- Growth factors (such as filgrastim) are allowed a minimum of 2 days after efti or pembrolizumab administration.
- Vaccination (e.g., influenza, COVID-19) with any non-live vaccine (e.g., vector-based, mRNA-based) is allowed if it takes place more than 3 days prior to or after any efti or pembrolizumab administration. Live attenuated vaccines cannot be used.
- Bisphosphonates and RANK-targeted therapy as clinically indicated.
- Subjects receiving opiates will be given preventive treatment for constipation and followed carefully.
- Inhaled or topical steroids.
- Acute surgery or elective (pre-planned) surgical procedures with non-oncological intent.

All concomitant medication will be recorded on the eCRF including all prescription, over-the-counter (OTC) products, herbal supplements, and i.v. medications and fluids. If changes occur during the study period, documentation of drug dosage, frequency, route, and date should also be included on the eCRF.

Prior chemotherapy (neoadjuvant or adjuvant, first line), targeted small molecule, anti-cancer monoclonal antibody or other systemic investigational drug therapy to treat the cancer disease including but not limited to are allowed in respective time windows defined in the inclusion and exclusion criteria and is to be recorded in the eCRF.

Prior high-dose chemotherapy requiring hematopoietic stem cell rescue or chemotherapy for metastatic disease is not permitted.

All concomitant medications received within 28 days prior to the first dose of study treatment and up to 30 days after the last dose of study treatment should be recorded. Concomitant medications administered 30 days after the last dose of study treatment should be recorded for SAEs and ECIs as defined in section 9.3 of the protocol.

The medical monitor should always be contacted to clarify and discuss the use of any concomitant therapies/procedures beforehand if not in line with the protocol.

## 3.5 Study Analysis Populations

There are 4 analysis populations defined for this study:

#### 3.5.1 Full Analysis Set

The Full Analysis Set (FAS) includes all assigned subjects who received at least one dose of study drug (i.e., one dose of either pembrolizumab or efti). This population will be the primary population for the analyzes of efficacy endpoints, demographics and baseline characteristics.

## 3.5.2 Evaluable Analysis Set (EAS)

The Evaluable Analysis Set (EAS) is a subset of the FAS and includes all subjects who received at least one dose of trial drug and has at least one evaluable post-baseline tumor assessment.


Prior Effective Date: 9th October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Subjects with best overall response as "NE (Not Evaluable)" or "NA (Not applicable)" will be excluded from the EAS population. This population will be the secondary population for efficacy analyzes based on overall response e.g., for ORR and PFS.

## 3.5.3 Per-Protocol Population

The Per-protocol (PP) population includes subjects in the FAS without major violation criteria (see Section 4.17). This population will not be used for any analyzes.

## 3.5.4 Safety Population

The safety set is defined analogously to the FAS and includes all assigned subjects who received at least one dose of study drug (i.e., one dose of either pembrolizumab or efti). This population will be the primary population for the analyzes of safety.

## 3.6 Withdrawn Subjects

Subjects should be withdrawn from the study if the subject:

- withdraws consent.
- is non-compliant with the study visits and procedures (refer to Section 7.4 of the protocol).
- becomes pregnant.

It is recommended that the Investigator attempts to perform an EOT visit evaluation if a subject withdraws consent during the treatment period.

The reason for subject withdrawal will be noted on the eCRF. The Investigator should attempt to follow withdrawn subjects until resolution of any adverse events, or at least 30 days after the last dose of study agent, or until completion of pregnancy whichever takes longer.

Upon withdrawal, no further dosing, or follow-up visits should be performed for these subjects. Investigators shall make reasonable attempts to contact lost-to-follow-up subjects for evaluation of OS.

Subjects may discontinue treatment other than for death, end of study, withdrawal of consent, lost to follow-up or (confirmed) progression, but remain on the study (e.g., PFS follow-up in case the subject has not progressed, otherwise OS follow-up) if:

- is non-compliant with the study treatments;
- the subject has clinically significant lab abnormalities or AEs (i.e., recurrent pneumonitis grade 2) that, in the Investigator's judgment, would preclude continued treatment;
- any other reason except withdrawal of consent;
- subject has attained a confirmed complete response and has been treated for at least 8 cycles receiving at least 2 cycles of pembrolizumab after the iCR was first declared.

The reason for treatment discontinuation will be noted and an end of treatment visit will be performed. The subjects should then continue with PFS and/or OS follow-up as applicable.

The data collected until the withdrawal of the subject will be used in the analysis.



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

The number of patients to be included in the study may be increased to achieve the expected number of patients with evaluable data for the primary objective analysis. Therefore, patients discontinued from study treatment due to SARS-CoV-2 infection before their on treatment radiological assessments including iRECIST assessment, were to be replaced.

### 3.7 Randomization

Not applicable as study is not randomized; subjects were assigned to the single treatment arm according to the indication as assessed during screening.

## 3.8 Blinding

Not applicable as study is a single treatment arm, open-label study.

## 3.9 Sample Size

The null hypothesis that the true response rate is [p0] will be evaluated against a one-sided alternative. In the first stage, [n1] subjects will be accrued. If there are [n1] or fewer responses in these [n1] subjects, the study will be stopped. Otherwise, [n-n1] additional subjects will be accrued for a total of [n]. The null hypothesis will be rejected if [n] or more responses are observed in [n] subjects. This design yields a type I error rate of [n] and power of when the true response rate is [n]. Calculations reveal that 17 subjects in the initial step and an additional 19 subjects, in total 36 subjects to be recruited into the study for the NSCLC first line and the other numbers as presented in the table below. Outcome of the calculation do not necessarily have to agree with the assumed proportions for the calculations  $[n]/N_1$  and  $[n]/N_1$  and  $[n]/N_2/N_1$  and  $[n]/N_1$  and  $[n]/N_2/N_2/N_2/N_3$  and  $[n]/N_1$  especially for such small sample numbers.

Mini-max results of this calculation were used for this clinical trial.

| Indication | Response rate p <sub>0</sub> | Alternative p <sub>1</sub> | r <sub>1</sub> | r <sub>2</sub> | Initial No of pts (n <sub>1</sub> ) | Add. No. of pts (n <sub>2</sub> ) | N <sub>total</sub> |
|---|---|---|---|---|---|---|---|
| NSCLC 1st line | 23% | CCI | 4 | CCI | 17 | 19 | 36 |
| NSCLC<br>2nd line | 7% | CCI | 1 | CCI | 23 | 13 | 36 |
| HNSCC | 15% | CCI | 2 | CCI | 18 | 19 | 37 |

The true response rates for 1<sup>st</sup> line NSCLC were extracted from Keynote-024 and Keynote-042 under consideration that for PD-1 all comers response rate will be lower. For 2<sup>nd</sup> line NSCLC there are no available publications for pembrolizumab alone in PD-1/PD-L1 refractory subjects, but due to the confirmation of progression it (p<sub>0</sub>) is considered close to 0% for pembrolizumab alone. The alternative (p<sub>1</sub>) of CCI was considered clinically relevant especially in comparison to available standard chemotherapy. For HNSCC relevant publications from Keynote-012 and Keynote-040 were used for p<sub>0</sub>.

Sample size calculations were performed using software R version 3.3.3 (2017-03-06), Package:

Kieser M, Wirths M, Englert S, Kunz CU and Rauch G (2017). "OneArmPhaseTwoStudy: An R Package for Planning, Conducting, and Analysing Single-Arm Phase II Studies." \_Journal of Statistical Software, \*81\*(8), pp. 1-28. doi: 10.18637/jss.v081.i08 (URL: <a href="http://doi.org/10.18637/jss.v081.i08">http://doi.org/10.18637/jss.v081.i08</a>).




| 1 Shoneor: Immilian S A S Protocol Nillmodr: | -002 (IMP321-<br>Keynote-PN798 |
|---|---|
|---|---|

For Part A an extension was anticipated based on the ORR of efti in combination with pembrolizumab as test group in a single arm design. The true ORR of monotherapy pembrolizumab in NSCLC 1<sup>st</sup> line is expected to be 23%, whereas a rate of color is expected for the test group (in case PD-L1 distribution is as expected from historical studies with ~70% <50% PD-L1expression). Using these assumptions with a power of color and a one-sided level of significance of color in this phase II trial, a sample size of 105 patients would be required for analysis. With a drop-out rate of 5%, a total of 110 patients need to be enrolled. With the 36 patients of stages 1 and 2, another 74 patients would be needed to be enrolled in total in this extension. This sample size is regarded sufficient to provide a reasonable precision for the estimate of ORR as basis for sample size considerations for further clinical studies.

Possible extensions of Part B and C will be introduced via substantial amendments.

Calculations were performed using PASS 2019 Power Analysis and Sample Size Software (2019). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass.

# 4 Statistical Methodology

## 4.1 Planned Analyzes

Baseline and demographic data will be summarized using the FAS population. Efficacy data will be summarized using the FAS and EAS populations (only final analysis). Safety data will be summarized using the safety population.

For continuous variables, data will be summarized by the number of subjects, mean, standard deviation, median, and minimum and maximum values. For categorical variables, data will be tabulated in frequency tables to display the number and percentage of subjects for each category.

Statistics will be displayed by part:

- Part A: NSCLC 1<sup>st</sup> line;
- Part B: NSCLC 2<sup>nd</sup> line:
- Part C: HNSCC 2<sup>nd</sup> line;

And by stage of inclusion. The stages will be derived as:

- Subjects include in Part A:
  - All subjects with Cycle 1 Day 1 (C1D1) date ≤ 30Jun19 should be included in stage 1.
  - All subjects with C1D1 date > 01Nov19  $\leq 30$ Sep20 should be included in stage 2.
  - All subjects with C1D1 date  $\geq$  01Oct20 should be included in stage 3 (extension).
- Subjects included in Part C:
  - All subject with C1D1 date  $\leq$  31Dec19 should be included in stage 1.
  - All subject with C1D1 date > 01Feb20 should be included in stage 2.
- Subjects included in Part B
  - All subject with C1D1 date  $\leq$  01Nov20 should be included in stage 1.
  - All subject with C1D1 date > 01Nov20 should be included in stage 2.



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

For some outputs overall (by stage for 1 part) or overall (all stages, all parts) will be generated.

#### **Notes:**

- Where a change from baseline is presented, if not specified in the footnote of the output, the results for baseline are defined as the last measurement obtained before the first dose of any study drug (efti or pembrolizumab, whichever occurs first); unscheduled assessment to be considered for determination of baseline only; the baseline is data collected at Cycle 1 Day 1 pre-dose for PK or TH1 biomarkers samples or at Screening for the gene expression.
- All data will be listed;
- The analyzes may be performed separately for each indication (dependent on availability of the results); if this is the case, only the column(s) for the relevant indication(s) will be included on tables;
- Separate clinical study reports (CSRs) may be written for each indication (dependent on availability of the results).

## 4.2 Timing of Analysis

Descriptive interim analyzes (including abbreviated reports, if needed) may be performed e.g., for the DMC meetings or when one stage of one part of the study is completed, which do not affect the analysis of the primary endpoint.

An initial descriptive interim analysis was performed with a data cut-off August 31, 2020. This interim analysis contained all subjects from stages who had completed enrolment (Part A and C). At least 90% of the subjects had a follow-up of  $\geq$ 18 weeks (e.g. 2 post baseline tumor stagings) at data cut-off.

The primary analysis was conducted once all patients were enrolled and had a follow-up of  $\geq$ 18 weeks (e.g., 2 post baseline tumor stagings) at data cut-off. The cut-off for the primary analysis was set July 1, 2022.

A follow up analysis (FU1) is planned to be conducted using the data cut-off date November 30, 2023. This analysis will have a minimum follow-up of 24 months, meaning that all subjects will have completed treatment.



This is an exploratory phase II umbrella trial. No formal hypothesis will be assessed.

Both DMC and the interim analysis do not affect the analysis of the primary endpoint. No adjustments for multiplicity are needed.

## 4.3 Disposition of Subjects

The number of subjects screened, assigned to treatment, in each analysis population, who completed/discontinued treatment and the reasons for any premature discontinuation from treatment will be presented by indication.




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

These analyzes will be produced in all screened subjects. Disposition will also be summarized by country and center.

## 4.4 Baseline and Demographic Characteristics

All baseline and demographic characteristics will be summarized by indication. This will include:

- Demographics: country, age, sex, race, ethnicity, male sexual status, female reproductive status, height, weight, body mass index (BMI), ECOG performance status, smoking status, duration of smoking at screening and number of cigarettes per day.
- Medical/surgical history: past medical history and concomitant diseases summarized by system organ class and preferred term.
- Cancer history:
  - o time since initial diagnosis (months), location (for HNSCC only), confirmed histological/cytological diagnosis, histology grade, tumor subtype, status of EGFR mutation (NSCLC only), status of ROS1 mutation (NSCLC only), status of BRAF mutation (NSCLC only), status of ALK translocation (NSCLC only), tumor stage at initial diagnosis, tumor stage at Screening; any metastatic disease (yes/no) and metastatic disease sites at screening (number and location of most frequent disease sites); brain metastases (Y/N); liver metastases (Y/N); HPV (HNSCC oropharyngeal only).

PD-L1 central assessment\_cat1 (by group: NSCLC: <1%, 1-49%, ≥50%, TPS, Not tested, Not evaluable; HNSCC: <1, 1-19, ≥20 CPS, Not Evaluable/Not Tested).

PD-L1 – derived central or local\_cat2 (by group: NSCLC: <1%, 1-49%, ≥50%, TPS, Not tested, Not evaluable; HNSCC: <1, 1-19, ≥20 CPS, Not Evaluable/Not Tested); priority for central PD-L1 and if not available take local data. HPV local assessment (Positive, Negative, and Not tested).

- History of HIV, HCV, HCV RNA, HBsAg.
- Active disease sites at baseline (any non-measurable lesions, Number of organs (site/location) affected by disease (target or non-target) and Site/Location.
- Other derived variables:
  - o Descriptive statistics for absolute counts of lymphocytes, neutrophils and monocytes, NLR at baseline.
  - Description Lactate dehydrogenase (LDH) abnormality normal (≤250 U/L) or abnormality high (>250 U/L).
  - Primary or secondary resistance (Part B only) definition in <u>Table 1</u>:
  - o Prior cetuximab (Prior Cetuximab, No Prior Cetuximab) Part C only.
  - Tumor Growth Kinetics Ratio numeric and categorical
  - Overall ADA (Positive/Negative).
  - Prior therapy Anti-PD-X



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

 Descriptive statistics of Maximum ALC Change from baseline up to and including Cycle 5 Day 1

- o Maximum ALC Change from baseline up to and including Cycle 5 Day 1 lloq
- o (<0.2/≥0.2 10^9/L)
- Baseline absolute lymphocyte count ( $<1.0/\ge1.0\ 10^9/L$ ).
- o Baseline NLR (<4.0/≥4.0)
- o NLR at Cycle 2 (<4.0/≥4.0)
- o TH1 biomarker relative change at Cycle 5 Day 1 Pre-DOSE (PCHG < or ≥40%)

Table 1: Definitions of primary and secondary resistance in advanced disease setting (acc. to SITC) (3)

| Resistance Type | Drug Exposure Requirement | Best Response |
|-----------------|---------------------------|---------------------------|
| Primary | ≥ 6 weeks | PD or SD for < 6 months |
| Secondary | ≥ 6 months | CR, PR, SD for > 6 months |

- Resistance is related to the last "Previous Systemic Anticancer Therapy Regimen" before efti and is related to the best response of their last therapy and how long they were on this treatment before progression.
  - Drug Exposure (months) = (Date of Progression Start Date of last previous Systemic Anticancer Therapy) +1.
- As per SITC the resistance is to be calculated for patients who had prior immunotherapy.
- For SD, check the duration between (Start Date/Time of Clinical Event Start Date/Time of last previous Systemic Anticancer Therapy.
- Active Disease site at baseline.

#### **Notes:**

- Age is recorded on the eCRF and will not be re-calculated.
- BMI will be calculated as weight (kg)/height<sup>2</sup> (m).
- Medical history is coded according to MedDRA version 21.1 or higher.
- Past medical history is defined as any medical/surgical history not marked as ongoing at time of screening.
- Concomitant diseases are medical/surgical history records marked as ongoing at the time of screening.
- Duration of Smoking at screening (Years) = (Years of stop date/Years of IC Years of start date). (Years of IC for current smokers).
- NLR = Neutrophil Count/Lymphocyte Count at baseline.

For Part A, the baseline characteristics are to be additionally presented by PD-L1 TPS (<1%, 1-49%,  $\ge$ 50%,  $\ge$ 1%). Note: this will be done for both central only and central or local.




## 4.5 Previous Anti-Cancer Therapy

- Any prior anti-cancer surgery (Y/N), [remark: from the eCRF 'Were there any prior cancer related surgeries = "Yes" and Intent of Surgery = "Palliative or Curative"]
- Any prior anticancer radiotherapy (Y/N);
- Any prior systemic anti-cancer therapy:
  - thereof chemotherapy (%)
    - thereof platinum (carboplatin, cisplatin or others) based therapy (%)
    - thereof targeting microtubules (e.g., paclitaxel, vinorelbine or others therapy (%)
    - thereof antimetabolites (5-FU, pemetrexed or others) therapy (%)
    - thereof DNA interacting (gemcitabine) therapy (%)
    - thereof other (%)
      - thereof drug name A
      - o thereof drug name B
  - thereof targeted therapy (%)
    - thereof anti-EGFR therapy (cetuximab or others) (%)
    - thereof other (%)
      - o thereof drug name A
      - o thereof drug name B
  - thereof immune checkpoint inhibitors (%)
    - thereof CTLA-4 based therapy
    - thereof PD-1/PD-L1 therapy (%)
      - o thereof PD-1 therapy
      - o thereof PD-L1 therapy
    - thereof other (%)
      - o thereof drug name A
      - thereof drug name B
  - any other systemic therapy (%)
    - o thereof drug name A
    - o thereof drug name B
- Any prior systemic therapy given with (neo-)adjuvant / curative intent; [remark: from the eCRF regimen name is not empty and Intention of therapy = "all except palliative"]
- Any prior systemic therapy given with palliative / symptomatic intent [remark: from the eCRF regimen name is not empty and Intention of therapy = "PALLIATIVE"]
- Last therapy prior to inclusion by intervention type:



| Sponsor: | Immutep S.A.S. | I Protocol Killmaner. | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

o radiotherapy alone

- o surgery alone
- o systemic therapy alone
- o combination of radiotherapy and/or surgery and/or systemic therapy [remark: Include all stop dates of radiotherapy, surgery and systemic therapy < inform consent date and select the last one;
- Last therapy prior to inclusion duration and best overall response
- Last therapy by intention of therapy:
  - o adjuvant/neoadjuvant
  - o curative
  - o palliative/symptomatic
- In case palliative / symptomatic by BoR
  - o PD, SD, PR, CR, unknown (The best response assessment linked to the last record in time is used.)
- In case last therapy contained systemic therapy split by:
  - Contained chemotherapy
  - Contained immune checkpoint inhibitor (ICI)
  - Contained targeted therapy
  - o Single agent therapy
  - Combination therapy
- Duration between any last anticancer intervention (i.e., surgery and/or radiotherapy) until date of informed consent (days)

[remark: inform consent date - last stop dates of radiotherapy, surgery+1]

• Duration between any last systemic anticancer therapy until date of informed consent (days)

[remark: inform consent date - last stop dates of systemic anticancer therapy+1]

• Number of prior systemic therapies for underlying cancer (0;1;2;>2)

#### **Notes:**

 Number of prior systemic therapies for underlying cancer: Consecutive records will be regarded as 1 line of therapy unless the time interval between the records exceeds 30 days. The eCRF grouping variable Regimen Number is used to identify same treatments lines.

### 4.6 Concomitant Medication

Prior medications comprise all therapies that were stopped prior to cycle 1 day 1. Medications used at study entry are defined as medication that started prior to the treatment period (cycle 1 day 1) and still ongoing at cycle 1 day 1. Concomitant medications are defined as medications that were started on or after cycle 1 day 1 until 28 days after end of treatment (last dose of any TPBS001 Version 6 CONFIDENTIAL Effective Date: 15<sup>th</sup> March 2017 (based on TPQA036 Version 2) Prior Effective Date: 9<sup>th</sup> October 2016



| Sponsor: | Immutep S.A.S. | I Protocol Killmaner. | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

study drug). Any medications started more than 28 days after last dose of any treatment are defined as post-treatment.

Incidence of prior medications, medications used at study entry and concomitant medication will be presented by indication, ATC name and preferred drug name (using the FAS). ATC name will be the highest coded ATC name (i.e., ATC level 4 if the medication is coded to level 4) (using the safety set).

Post-treatment medications will be listed only.

Where a medication start date is partially or fully missing, and it is unclear as to whether the medication is prior, used at study entry, concomitant or post-treatment, it will be assumed that it is concomitant.

#### **Notes:**

• Medications are coded using WHO Drug dictionary, version SEP2018 or higher.

## 4.7 Concomitant Procedures

Concomitant procedures will be assessed, starting from cycle 1 day 1 until 28 days after end of treatment (last dose of any study drug). Concomitant procedures will be summarized by system organ class and preferred term (using the safety set).

#### **Notes:**

• Procedures are coded according to MedDRA version 21.1 or higher.

## 4.8 Exposure and Compliance

For efti and pembrolizumab separately, exposure is defined as:

- Exposure (weeks) =  $\frac{\text{date of last dose} \text{date of first dose} + 1}{7}$ .
- Follow-up time (months) = (date of last available information in the study date of first dose + 1)/30.4375.

Note: Subjects who miss more than a total of 3 injections of efti or 2 infusions of pembrolizumab within the first 8 cycles or a total of more than 5 doses of efti or pembrolizumab until cycle end of combination treatment (end of cycle 18) will be regarded as treatment non-compliant. Subjects will need to end the treatment as per protocol.

For efti, the following summaries will be produced:

- Descriptive summary of exposure (weeks);
- Descriptive summary of exposure (months);
- Descriptive summary of the total number of doses received;
- Number and percentage of subjects with 1, 2 or > 2 treatment delay/interruptions and number and % of pts permanently discontinued
- Number and percentage of subjects with 1, 2, 3 or >3 missed doses within the first 8 cycles;


SAP Version 3, Final


Effective Date: 15th March 2017

31Jan2024



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Number and percentage of subjects with 1, 2, 3, 4, 5 or >5 missed doses during the whole combination treatment period;

- Number and percentage of compliant and non-compliant subjects as described above;
- Number and percentage of subjects withdrawn from treatment due to non-compliance.

For pembrolizumab, the following summaries will be produced:

- Descriptive summary of exposure (weeks);
- Descriptive summary of exposure (months);
- Descriptive summary of the total number of doses received;
- Number and percentage of subjects with 1, 2 or >2 treatment delay/interruptions and number and % of pts permanently discontinued
- Number and percentage of subjects with 1, 2 or >2 missed doses within the first 8 cycles;
- Number and percentage of subjects with 1, 2, 3, 4, 5 or >5 missed doses during the whole combination treatment period;
- Number and percentage of compliant and non-compliant subjects as described above;
- Number and percentage of subjects withdrawn from treatment due to non-compliance.

Exposure and compliance will also be described for efti and pembrolizumab combined, the definitions provided above will apply. First/last dose refers to efti or pembrolizumab whichever one come first.

In case there is a next visit treatment entered in row (i.e., no gap in numbering of visits), no matter how long after previous treatment, which should be regarded as delay/interruption and not missed dose.

## 4.9 Efficacy Analysis

iRECIST and RECIST 1.1 are used for the tumor evaluation see Section 8.1 of the protocol (efficacy assessment). iRECIST is based on RECIST 1.1 but adapted to account for the unique tumor response seen with immunotherapeutic drugs.

All efficacy analyzes are based on local Investigator assessments. The interim analysis, primary and FU1 analyzes have also been evaluated by a Blinded Independent Central Reviewer (BICR).

Efficacy analyzes will be performed for each part (A, B or C) of the study independently. It may be split by stage for ORR.

#### 4.9.1 Primary Endpoint Analysis

### 4.9.1.1 Primary Efficacy Endpoint: iORR according to iRECIST

The primary endpoint, iORR, is defined as the proportion of subjects with a best objective response (iBOR) of complete response (iCR) or partial response (iPR) according to iRECIST.

TPBS001 Version 6 (based on TPQA036 Version 2) CONFIDENTIAL



| Sponsor: | Immutep S.A.S. | I Protocol Killmaner. | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

The iBOR is the best response as determined by the Investigator (and BICR, if assessed) between the date of assignment and date of objective measurement of iUPD or iCPD by iRECIST, the date of subsequent therapy or date of lost to follow-up, whichever comes first.

The overall responses at each visit are used to determine the iBOR. iBOR will be assigned using the following categories (from best to worst responses): complete response (iCR), partial response (iPR), stable disease (iSD), unconfirmed disease progression (iUPD), confirmed disease progression (iCPD) or not evaluable (NE) at each timepoint.

iSD can only be assigned as iBOR if the patient has a best response of iSD that is at least 6 weeks after the date of treatment assignment (on or after study Day 43, 42 days after date of first dose of study treatment). If the patient had no subsequent post-baseline data, then the iBOR will be NE.

For BICR results iBOR of "Non-iCR/Non-iUPD" should be considered "iSD" for programming and will be included in the iDCR.

#### **Unconfirmed iBOR:**

Defined as the iBOR recorded during the observation period defined in Section 4.9.1.1.

#### **Confirmed iBOR:**

Applicable only for subjects with an iBOR of iCR or iPR, a response may be considered confirmed if observed at subsequent radiological assessments at least 4 weeks apart and there are no assessments with an overall response of iSD or iUPD between the 2 assessments. Alternatively, an iBOR of iCR that does not meet the criteria for confirmed iCR may still meet the criteria of confirmed iPR if there is a response of iPR that is confirmed with an overall response of iCR at least 4 weeks apart and there are no assessments with an overall response of iPR if the overall response of iPR is confirmed with an overall response of iPR at least 4 weeks apart and there are no assessments are not assessments

See <u>Table 2</u> below for the derivation of confirmed iBOR when iCR or iPR is believed to be the iBOR.




Table 2: iBOR when confirmation of iCR and iPR is required

| Table 2. IDOK when confir mation of iCK and if K is required | | | |
|---|---|---|---|
| Response:<br>First Time<br>Point | Subsequent Time<br>Point | BOR | Also Requires |
| iCR | iCR | iCR | Normalization of tumor markers. All tumor nodes <10 mm. |
| iCR | iPR | iSD, iUPD or iPR (see comment*) | |
| iCR | iSD | iSD provided minimum criteria for iSD duration met, otherwise, iUPD | |
| iCR | iUPD | iSD provided minimum criteria for iSD duration met, otherwise, iUPD | |
| iCR | NE | iSD provided minimum criteria for iSD duration met, otherwise NE | |
| iPR | iCR | iPR | |
| iPR | iPR | iPR | |
| iPR | iSD | iSD | |
| iPR | iUPD | iSD provided minimum criteria for iSD duration met, otherwise, iUPD | |
| iPR | NE | iSD provided minimum criteria for iSD duration met, otherwise NE | |
| NE | NE | NE | |

<sup>\*</sup> If iCR is truly met at first time point, then any disease seen at a subsequent time point, even disease meeting iPR criteria relative to baseline, makes the disease iUPD at that point (since disease must have reappeared after iCR). Best response would depend on whether minimum duration (at least 6 weeks after start of treatment) for iSD was met.

For each part (and stage dependent on the time of analysis) separately and for both the FAS and EAS populations, iORR will be summarized by binomial response rate with two-sided 95% exact confidence intervals (CIs) using the Clopper-Pearson method.

### 4.9.2 Secondary Endpoints Analyzes

All secondary analyzes will be performed descriptively and based on local assessments and BICR, if assessed.

#### 4.9.2.1 Secondary Efficacy Endpoint: ORR According to RECIST 1.1

ORR follows the same definition used by iRECIST in Section 4.9.1.1, using however the RECIST 1.1 criteria to assess responses (4).

ORR, per RECIST 1.1, is defined as the proportion of subjects with a best objective response (BOR) of complete response (CR) or partial response (PR).

The overall responses at each visit are used to determine the BOR. BOR will be assigned using the following categories (best to worst): CR, PR, SD, PD and NE.

The principles of unconfirmed and confirmed responses (for BOR PR or CR) are as previously described per iRECIST. Similar analyzes will be conducted for ORR as described for the primary endpoint iORR.


Prior Effective Date: 9<sup>th</sup> October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

# 4.9.2.2 Secondary Efficacy Endpoint: Disease Control Rate (DCR) According to iRECIST and RECIST 1.1

iDCR is defined as the percentage of subjects achieving an unconfirmed iCR, iPR or iSD (iSD duration from C1D1 lasts at least 6 weeks) as iBOR.

iDCR will be analyzed using the same methods specified for iORR.

DCR (per RECIST 1.1) will be analyzed using the same methods specified for iDCR.

# 4.9.2.3 Secondary Efficacy Endpoint: Progression Free Survival (PFS) According to iRECIST and RECIST 1.1

iPFS is defined as the time from the date of first treatment (C1D1) to the date of first documentation of disease progression per iRECIST (iUPD, except when there is a subsequent timepoint with iSD, iPR or iCR and no iCPD in between) or date of death due to any cause, whichever occurs first:

PFS (months) =

 $\underline{\textit{Date of First Documented Progression/Death/Censoring Date -Date of start of treatment (C1D1) + 1}}_{30.4375}$ 

For subjects without progression or death, iPFS will be censored as described in Table 3.

The iPFS rate at 3, 6, 12, 18, 24, 36 and 48 months and corresponding 95% CIs will be estimated using the Kaplan-Meier method. The total number of patients who experienced the event and number of patients censored will also be reported. iPFS will also be displayed graphically using a Kaplan-Meier plot.

As per iRECIST guidelines, disease progression can be confirmed by the site 4–8 weeks from the scan showing iUPD if the subject is clinically stable. This may correspond to the next visit in the original visit schedule. The assessment of the subsequent confirmation imaging proceeds in an identical manner, with possible outcomes of iCPD, iUPD, and iSD/iPR/iCR. Subjects who have unconfirmed disease progression and are clinically stable can continue treatment until progression is confirmed.

PFS will be summarized similarly to iPFS based on RECIST 1.1.

Table 3: Censoring Rules for PFS for RECIST and iRECIST

| Situation | Date of Progression or Censoring | Outcome |
|---|---|---|
| Death or disease progression between planned radiological assessments | Date of death or first radiological assessment showing disease progression, whichever occurs first | Progressed |
| Death before first radiological assessment | Date of death | Progressed |
| No baseline or post-baseline radiological assessments | Start date of first treatment | Censored |
| New anticancer treatment started<br>before documentation of disease<br>progression or death | Date of last radiological assessment prior to the start of non-protocol anticancer treatment | Censored |
| Death or progression after one missed radiological assessment | Date of missed radiological assessment visit | Progressed |



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

| Situation | Date of Progression or Censoring | Outcome |
|---|---|---|
| Death or progression after two or | Date of last radiological assessment visit | |
| more consecutive missed radiological | without documentation of disease | Censored |
| assessments | progression that is before the missed visit | |
| Two consecutive missed, scheduled | Date of last radiological assessment | Censored |
| radiological assessment (+ windows) | Date of last radiological assessment | |
| Alive and without documentation of | Date of last radiological assessment | Censored |
| disease progression | Date of last radiological assessment | |
| Additional censoring rules specific for iRECIST handling of PD assessments | | |
| If progression = iUPD and iUPD is | Date of the first radiological assessment | |
| identified as the last iRECIST | of iUPD in sequence leading to a final | Progressed |
| assessment (not confirmed) | iUPD result <sup>2</sup> | |
| If progression = iCPD and the iUPD | Date of the first radiological assessment | |
| then iCPD are consecutively | of iUPD in sequence leading to a final | Progressed |
| confirmed | iCPD result <sup>2</sup> | |
| If progression = iUPD* but neither | | |
| confirmed nor identified as PD for | Date of last radiological assessment | Censored <sup>2</sup> |
| subsequently performed iRECIST | Date of fast faulological assessificili | |
| assessments | | |

<sup>&</sup>lt;sup>1</sup> May be only one or multiple, consisting of a pattern of repeated iUPD tumor assessment results.

<u>Table 4</u> below describes examples of censoring rules for iPFS using iRECIST Guidelines.

Table 4: Example of censoring rules for iPFS using iRECIST

| Date 1 | Outcome 1 | Date 2 | Outcome 2 | Date 3 | Outcome 3 | Used for PFS per iRECIST |
|---|---|---|---|---|---|---|
| 01.01.2020 | iUPD | 15.03.2020 | iPR | Pt left study | NA | No event → censored with 15.03.2020 |
| 01.01.2020 | iUPD | pt left study | NA | NA | NA | PD event 01.01.2020 |
| 01.01.2020 | iUPD | 15.03.2020 | iPR | 25.06.2020 | iUPD | PD event 25.06.2020 |
| 01.01.2020 | iUPD | 15.03.2020 | iCPD | | | PD event<br>01.01.2020 |

# 4.9.2.4 Secondary Efficacy Endpoint: Duration of Response (DoR) according to iRECIST and RECIST 1.1

The response will be further evaluated by iDoR based on iRECIST. iDoR is calculated only for subjects with a confirmed iBOR of iCR or iPR up to an objective documentation of progression or death, whichever occurs first.


<sup>&</sup>lt;sup>2</sup> Censoring may also be required per rules above.


| Sponsor: | Immutep S.A.S. | Protocol Nilimper | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

 $iDoR (months) = \frac{Date \ of \ First \ Disease \ Progression/Death/Censoring \ date - Date \ of \ First \ iCR \ or \ iPR \ + 1}{30.4375}$ 

Progression and censoring dates for iDoR are determined the same way as iPFS (see Table 3).

For subjects who receive subsequent anticancer therapy prior to objective disease progression, iDoR will be censored at the date of the last tumor assessment date prior to the date of subsequent therapy.

For each indication separately and for the FAS population, iDoR will be summarized using the Kaplan-Meier method. The median time to event will be calculated along with 95% CIs using the Kaplan-Meier method. Mean (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles and minimum and maximum values will also be presented. In addition, the proportion of responders still in response at 3, 6, 9, 12, 18 and 24 months will be presented.

iDOR will also be displayed graphically using a Kaplan-Meier plot.

DoR will be presented in the same way as iDoR based on RECIST 1.1.

# 4.9.2.5 Secondary Efficacy Endpoint: Time to Response (TTR) According to iRECIST and RECIST 1.1

iTTR will be evaluated for the subset of patients categorized as confirmed responders for the assessment of iORR.

iTTR is defined as the time from start of treatment (C1D1) to first iCR or iPR response.

$$iTTR (months) =$$

$$\underline{Date \ of \ First \ iCR \ or \ iPR \ - Date \ of \ start \ of \ treatment \ (C1D1) \ + 1}}{30.4375}$$

For each indication separately and for the FAS population, iTTR will be summarized using descriptive statistics including mean (SD).

TTR will be presented in the same way as iTTR based on RECIST 1.1.

#### 4.9.2.6 Overall Survival (OS)

All subjects in the trial will be followed up for survival until death, end of the trial, withdrawal of consent, or loss to follow-up, whichever of these occurs first.

OS is defined as the time from the start of the treatment (C1D1) to the date of death due to any cause. For subjects still alive at the time of analysis, OS will be censored at the date the subject was last known to be alive.

$$OS (months) = \frac{Date \ of \ Death/Last \ Known \ to \ be \ Alive - Date \ of \ Start \ of \ Treatment \ (C1D1) + 1}{30.4375}$$




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Date of Last Known to be Alive is the last date with available information for a subject in the study.

For each separate indication, using the FAS population, OS will be summarized using the Kaplan-Meier product-limit method. The median time to event will be calculated along with 95% CIs using the Kaplan-Meier method. Mean (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles and minimum and maximum values will also be presented. The OS rate at 3, 6, 12, 18, 24, 36 and 48 months and corresponding 95% CIs will also be estimated using the Kaplan-Meier method.

OS will also be displayed graphically using a Kaplan-Meier plot.

## 4.9.3 Exploratory Efficacy Endpoint Analyzes

## 4.9.3.1 Exploratory Efficacy Endpoint: Circulating biomarkers

Plasma samples will be collected prior to dosing on Day 1 of Cycles 1, 5, 9, 13, end of combination (EOC) therapy and at EOT to assess for Th1 biomarkers (IFN-γ, CXCL10/IP10, CXCL11/iTAC) at the central laboratory (Charles River Laboratories). Results with < LLOQ or > ULOQ are set at the LoQ value for analysis purposes and can be identified in the listing.

In the subset of subjects with PK assessment, Th1 biomarkers may be additionally assessed in samples collected at selected time points after dosing with efti at cycle 1, cycle 5 and cycle 9.

Available results for each circulating TH1 biomarker of interest will be listed and summarized by indication, visit and time point (if applicable) using the FAS. Descriptive statistics (including quartiles) will be reported for absolute values and absolute and percentage change from baseline calculated as follows,

Percentage Change = 100\* (Value at the visit – Value at Baseline)/Baseline value

#### 4.9.3.2 Exploratory Efficacy Endpoint: Gene Expression Profiling

Whole blood samples were collected in PaxGene tubes for gene expression profile (GEP) analysis at the central laboratory (Covance/Labcorp, Indianapolis) prior to dosing at screening and cycle 5 day 1.

GEP analysis was done separately and is not part of this SAP.

A separate analysis report will be developed and will be included as appendix to the CSR.

# 4.9.3.3 Exploratory Efficacy Endpoint: Co








CCI

# CCI

analyzed on FAS and EAS population.

## 4.9.4 Other Exploratory Endpoints

## 4.9.4.1 Exploratory Endpoint: Tumor PD-L1 Expression

Archival tumor material or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated was provided by subjects on a mandatory basis. PD-L1 expression was centrally analyzed by Covance, Geneva. Results will be displayed with an overall score CPS (HNSCC, Part C) and TPS (NSCLC, Parts A and B). Available locally obtained results will also be included.

PD-L1 expression status in tumor tissue will be provided as by subject including subject ID, stage and part of the trial, score and type of score (TPS/CPS) for centrally and locally obtained results. A pre-defined cutoff will be used to determine PD-L1 expression status (see Section 4.4).

Centrally assessed PD-L1 results (from Covance lab) should be primarily used. For subjects whose PD-L1 result was found not evaluable by the central lab, the PD-L1 result assessed in the local laboratory will be used. Two different populations will be used for efficacy analysis:

- 1. Central only
- 2. Central or local (meaning that for each patient where central was not available but local the local result will be used)

The data for local PD-L1 is collected in the eCRF as numerical and as categorical. It may happen that the numerical value is empty when the categorical value is negative, i.e., <1% for TPS. For the analysis and consistency, the derived categorical data which contains the items "<1%; 1-49% and  $\geq$ 50%, will be created by considering these data in the item the category "<1%". If numerical value is empty and categorial is "negative" then the derived variables will take a value "<1%" for categorial and 0 for numerical.

## 4.9.4.2 Exploratory Endpoint: Immunogenicity

Autoantibodies such as antimitochondrial antibodies, rheumatoid factor, antithyroid (antithyroglobulin) antibodies, and antinuclear antibodies will be evaluated at the local laboratory at cycle 1 day 1, cycle 9 day 1, EOC and EOT.

The formation of anti-drug antibodies (ADA) against efti and their neutralizing capacity (Neutralizing Antibody, Nab) will be assessed at the central laboratory (Charles River Laboratories) in blood samples collected at cycle 1 day 1, cycle 2 day 8, cycle 3 day 15, cycle 5 day 1, cycle 9 day 1, cycle 13 day 1, EOC prior to dosing and at the EOT visit.

Results for each immunogenicity parameters will be summarized by indication and per visit (including C1D1) as % positive, negative or non-tested samples (using the FAS) and as descriptive statistics for ADA-titer and Nab-titer (including quartiles). For ADA and Nab,




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

overall results will also be presented by considering the results of all post-baseline visits, for the categorical variable (i.e., ADA positive/negative or Nab positive/negative), if at least one post baseline timepoint (visit) is positive then subject need to be reported as positive; for the numeric values, the maximum value of all post-baseline visits will be considered for overall (peak ADA-titer or peak Nab-titer).

## 4.10 Pharmacokinetic Analysis

Pharmacokinetics analysis will be provided to Immutep by PhinC development according to analytical plan using the plasma concentration of LAG-3 results generated by Charles River Laboratories Saint Nazaire.

PK analysis was done separately and not part of this SAP.

A PK analysis report will be developed by PhinC and included as appendix to the CSR.

# 4.11 Subgroup Analysis

The subgroups listed below will be analyzed for ORR, PFS (per iRECIST and RECIST 1.1) and OS. DOR (per iRECIST and RECIST 1.1 is required for selected subgroups, defined in <u>Table 5</u>. All subgroup analysis will be done based on investigator assessment for the FAS population. The details for each subgroup and part are listed in <u>Table 5</u>.

The following subgroups will be analyzed:

- PD-L1 status (central only and central or local):
  - PD-L1 NSCLC (Part A)
    - Negative (<1% TPS); TPS 1-49%; TPS ≥50% and Positive (≥1% TPS).
  - PD-L1 NSCLC (Part B)
    - Negative (<1% TPS); TPS 1-49%; TPS <50%; TPS ≥50% and Positive (≥1% TPS).
  - PD-L1 HNSCC (Part C)
    - Negative (<1 CPS); 1-19 CPS;  $\geq$ 20 CPS; <20 CPS and Positive ( $\geq$ 1 CPS).

Effective Date: 15<sup>th</sup> March 2017 Prior Effective Date: 9<sup>th</sup> October 2016

- Sex:
  - Male
  - Female
- Smoking Status:
  - Never
  - Former
  - Current
  - Former + current
- Age:
  - <65 years
  - ≥65 years
- ECOG Performance Status at screening:
  - (
  - 1
- Overall ADA (see Section 4.9.4.2):




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Positive

- Negative
- Region:
  - Spain
  - Non-Spain
- Tumor Type (Part A only):
  - Squamous
  - Non-Squamous

[remark: this information will be derived from the eCRF 'Cancer History Log Form', subject with tumor type or sub-type "Squamous Cell Carcinoma" will be included in the item Squamous]

- Resistance (Part B only):
  - Primary
  - Secondary
- Prior cetuximab (Part C only):
  - Prior cetuximab
  - No prior cetuximab
- HPV status (for Part C subjects with primary oropharyngeal tumors only):
  - Positive
  - Negative
  - Not Done/Not tested

[Remark: this information will be derived from the eCRF 'Histology Cytology assessment details Log Form' HNSCC: Status of HPV item (Positive=yes, Negative=no, Not Done/Not tested].

The subgroup analysis for this category will be performed only if at least 10 subjects are identified with positive HPV.

- Prior Therapy (Part B only; please see derivation rules provided in Appendix 5.6.2):
  - Anti-PD-X-based treatment + chemo
  - Anti-PD-X-based therapy alone or + ICI
- Maximum Absolute Lymphocyte count (ALC) change (all parts):
  - Max. ALC on treatment (any post study treatment initiation value till C5D1 versus baseline (C1D1 or Screening in case baseline is not applicable):
    - 1.  $<0.2\ 10^9/L$ ;
    - 2.  $\geq 0.2 \ 10^{9}$ L.

Table 5. Summary of required analyzes per subgroup (Investigator only)

| Subgroup | Part A | Part B | Part C |
|----------------------|-------------------|--------|--------|
| PD-L1 central only | | | |
| <1%<br>1-49%<br>≥50% | ORR, PFS, DoR, OS | NA | NA |
| ≥1% | | | |
| <50% | | | |




| | <u>, </u> | | |
|---|---|---|---|
| <1<br>1-19<br>≥20 | NA | NA | ORR, PFS, DoR, OS |
| >1 | | | |
| <20 | | | |
| PD-L1 central or local | | | |
| <1%<br>1-49%<br>≥50% | ORR, PFS, DoR, OS | NA | NA |
| ≥1% | | | |
| <1%<br>1-49% | NA | ORR, PFS, OS | NA |
| <50%<br>≥1% | | | |
| ≥50% | | | |
| <1<br>1-19<br>≥20 | NA | NA | NA |
| <20 | | | |
| Sex | ORR, PFS, OS | ORR, PFS, OS | ORR, PFS, OS |
| Smoking status | | | |
| Former or current Never | ORR, PFS, OS | ORR, PFS, OS | NA |
| Former<br>Current<br>Never | NA | NA | ORR, PFS, OS |
| Age | ORR, PFS, OS | ORR, PFS, OS | ORR, PFS, OS |
| ECOG | ORR, PFS, OS | ORR, PFS, OS | ORR, PFS, OS |
| Overall ADA | ORR, PFS, OS | ORR, PFS, OS | ORR, PFS, OS |
| Region | ORR, PFS, OS | ORR, PFS, OS | ORR, PFS, OS |
| Tumor type | ORR, PFS, DoR, OS | NA | NA |
| Resistance | NA | ORR, PFS, OS | NA |
| Prior cetuximab | NA | NA | ORR, PFS, OS |
| HPV status | NA | NA | ORR, PFS, OS |
| Prior therapy | NA | ORR, PFS, OS | NA |
| ALC change | ORR, PFS, OS | ORR, PFS, OS | ORR, PFS, OS |
| Note: ORR, PFS and DoR to be | presented by both iRECIST ar | nd RECIST 1.1. | |




| Sponsor: Immutep | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|
|---|---|---|

## 4.11.1 Efficacy (Investigator only) by ALC change under therapy

KM for OS and PFS (iRECIST and RECIST 1.1) based on "Maximum ALC Change from baseline up to Cycle 5 Day 1– cat" will be presented in table and figure by part.

Boxplot of Max ALC Change will be displayed for confirmed iBOR (iCR + iPR vs Others) and iDCR (iCR+ iPR+ iSD vs Others) by part.

## 4.11.2 Overall Survival (OS) by Response (Investigator assessment only)

OS will be summarized by best overall response according to iRECIST per local assessment as described below and will be presented in a table and figures.

#### Part A:

- Confirmed iCR + iPR;
- Unconfirmed iPR + iSD;
- iUPD/iCPD + iNA/iNE

## Part B:

- Confirmed iPR + iSD;
- iUPD/iCPD + iNA/iNE;

## Part C:

- Confirmed iCR + iPR;
- Unconfirmed iPR + iSD + iUPD/iCPD + iNA/iNE.

## **4.12 Tumor Growth Kinetics**

Tumor growth kinetics (TGK) are to be calculated for each subject in Part B whose identical target lesions have been tracked from pre- to post-baseline by local assessment and BICR.

Table 6. Example to determine which patients should be included for TGK analysis

| Reference scan target tumor lesions | Post-baseline target tumor<br>lesions | Patient to be included? |
|---|---|---|
| Lung (left lower lobe lung nodule) | Lung (left lower lobe lung nodule) | Yes |
| Lung (lower right lobe) Lymph node (right hilar) | Lung (lower right lobe) Suprarenal gland (left adrenal) | Yes- but only including measurements from lung (lower right lobe) |
| Lung (left upper lobe) | Lung (left supra clavicular node) | No |

The list of patients and their lesions which should be part of tumor growth kinetics analysis in Part B are indicated in the appendix Section 5.6.1.

This calculation is based on a ratio comparing pre-treatment tumor behavior to the on-study tumor behavior (5). The following definitions are part of this calculation:




T1: date and time of confirmatory pre-baseline scan\*

TPRE: date and time of reference scan

T0: date and time of baseline

TPOST: date and time of best post-baseline scan

S1: sum of the largest diameter of target lesions at confirmatory pre-baseline scan\*

SPRE: sum of the largest diameter of target lesions at reference scan

S0: sum of the largest diameter of target lesions at baseline

SPOST: sum largest diameter of target lesions of best post-baseline scan (best post baseline = smallest post baseline value).

\*If the confirmatory pre-baseline scan data is not available for any reason, then the initial progression pre-baseline scan may be used (ensuring that the same lesions are followed).

Using the above definitions, TGKPRE is calculated as the difference of the sum of the largest diameters of the target lesions (according to iRECIST or RECIST 1.1) per unit of time (months) between pre-baseline and baseline imaging:

$$TGKPRE = (S1-SPRE) / (T1-TPRE).$$
  
 $TGKPOST(=(SPOST-S0) / (TPOST-T0).$ 

The final calculation of TGK ratio (TGKR) is defined as the ratio,

Shrinkage= TGKR<0

Deceleration= 0<TGKR<1

Acceleration=TGKR≥1

To present a figure on tumor dynamics, each applicable patient is to have three points:

- 1. Reference scan: Months from baseline (x-axis), % change from baseline (y-axis)
- 2. Baseline: Months from baseline (x-axis), % change from baseline (y-axis), i.e. (0.0)
- 3. Best post-baseline scan: Months from baseline (x-axis), % change from baseline (y-axis)

These 3 points are to be joined by a line that is color coded by the patient's TGKR.

Shrinkage= green

Deceleration= orange

Acceleration= red

TGK ratio will be derived and summarized as numeric and categorical parameter as described above. The corresponding figure will also be presented.

Tumor growth kinetics will also be analyzed using the data from BICR. Same tabulation and figure as described above will also be repeated using BICR data.

## 4.13 Safety Analysis

The safety endpoints of this study are the frequency, severity and duration of AEs, SAEs, ECIs and abnormalities in vital signs, physical examination, 12-lead ECG and safety laboratory and urine assessments.


Prior Effective Date: 9th October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

### 4.13.1 Adverse Events

An AE summary table will include treatment-emergent adverse events (TEAE; i.e., AEs with onset dates on or after the first dose of study drug regardless of causality), serious TEAEs, ECIs, TEAEs related to efti, TEAEs related to pembrolizumab, fatal TEAEs (i.e. AE grade 5 and/or AE outcome death), TEAEs leading to temporary and permanent discontinuation of treatment (each treatment separately) and discontinuation from study treatment, TEAEs according to worst severity and combinations of previously mentioned type of AEs. For each parameters causality information will be shown as specified below.

The number and percentage of subjects with at least 1 TEAE will be tabulated by preferred term and system organ class. For these tabulations, the number of subjects (i.e., subjects with multiple events will be counted only once per preferred term) and the number of events (i.e., except for by severity tabulations) with that particular TEAE are presented. For severity tabulations highest grades will be shown. Similar tables will be produced for serious TEAEs, fatal TEAEs, TEAEs leading to permanent discontinuation of treatment, discontinuation from study and events of clinical interest. The previously mentioned type of TEAEs might also be presented in combination with treatment-relatedness.

AEs will also be tabulated by severity and relationship to each study drug. At each level of tabulation, the event with the highest level of severity or strongest drug relationship will be presented. Possibly related and Related assessment in the clinical database translates to Related in the outputs. Causality information will be shown as (1) related to efti, (2) related to pembro, (3) related to trial treatment (i.e., efti and/or pembro) and (4) regardless of relationship (as applicable).

All AEs will be listed. In addition, detailed listings will be provided for subjects who die, experience a SAE, or discontinue the study because of an AE. These listings will include age, duration of follow up, number of doses received, and time since last dose of pembro and efti, respectively. Events with a time of onset within 24 hours from time of most recent efti injection will be flagged (using the flag: 24-hr) if the event time is missing and event date is the same as date of efti injection the event will be flagged.

Non-treatment emergent events (starting prior to exposure to study treatment) will be included in the subject listings and flagged but will not be included in the above summaries. Where an AE start date is partially or fully missing, and it is unclear as to whether the AE is treatment emergent, it will be assumed that it is.

AEs with a coded PT meeting the broad Standardized MedDRA Query (SMQ) "Hypersensitivity" will be listed. AEs occurring within 24 hours from most recent efti injection will be flagged.

AEs with a coded preferred term meeting the broad MedDRA SMQ "Extravasation events (injections, infusions and implants)" and including PT "Injection site reaction", at least possibly related to efti and/or adverse events with indication "local injection site reaction in the clinical database will be listed.

Patients with a recurrent adverse reaction (i.e., adverse reactions at least possible related to efti) indicating systemic inflammatory response with onset date within 24 hours after efti injection will be listed.

Patients with adverse reaction indicating immune-related adverse event will be listed.

TPBS001 Version 6 CONFIDENTIAL Effective Date: 15<sup>th</sup> March 2017 (based on TPQA036 Version 2) Prior Effective Date: 9<sup>th</sup> October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Non-treatment emergent events (starting prior to exposure to study treatment) will be included in the subject listings and flagged but will not be included in the above summaries. Where an AE start date is partially or fully missing, and it is unclear as to whether the AE is treatment emergent, it will be assumed that it is.

Systemic inflammatory response will be summarized and listed. Terms to be used for selection include chills, cytokine release syndrome, feeling cold, feeling hot, influenza like illness, malaise, myalgia, post-procedural complication, pyrexia.

Based on the selection above,

- ✓ A listing will be created with all events which are within 24 hrs from efti intake and are a matching term even if unrelated to efti, and even if only one event per patient.
- ✓ A table who include only the patients who have at least two such of events and both are related to efti, and both have start date 24 hrs from the intake of efti OR one matching term the verbatim of which includes "intermittent" (or variation thereof) and is related to efti and start is w/in 24 hrs from intake of efti

Patients with adverse reaction indicating immune-related adverse event will be listed.

Immune-Related Adverse Events (irAEs) will be summarized per groups term and pertaining PTs and per severity grades and listed. Grouping (in bold) and preferred MedDRA terms to be used for selection are listed in the Table 7:

Table 7: irAEs (Adverse reactions – at least possibly related to either pembro and/or efti)






| irAEs (adverse reactions – at least po | ssibly related to either peml | bro and/or efti) |
|---|---|---|
| | | Preferred Terms |
| | | ca |
| Colitis | | |
| | | CCI |
| | | CCI |
| Severe Skin Reactions (i.e., ≥gr 3) | | |
| Severe Skiii Reactions (i.e., Egr 3) | | |
| Hepatitis | | |
| Thyroiditis | | |
| Advanal Insufficionar | | |
| Adrenal Insufficiency | | |
| TPBS001 Version 6 | CONFIDENTIAL | <mark>ccl</mark><br>Effective Date: 15" March 201. |
| (based on TPQA036 Version 2) | | Prior Effective Date: 9th October 2016 |



| irAEs (adverse reactions – at least possibly related to either pembro and/or efti) | |
|---|---|
| Pre | eferred Terms |
| CCI | |
| Hypophysitis | |
| CCI | |
| Nephritis | |
| Myositis | |
| Pancreatitis | |
| Type 1 Dich stee Mallitus | |
| Type 1 Diabetes Mellitus | |
| CCI | |
| Uveitis | |
| CCI | |




| irAEs (adverse reactions – at least possib | ly related to either pembro and/or efti) |
|---|---|
| | Preferred Terms |
| | CCI |
| | COI |
| Sarcoidosis | |
| Sarcoldosis | CCI |
| 3.5 | 001 |
| Myocarditis | |
| | CCI |
| | <u> </u> |
| Encephalitis | |
| | CCI |
| Guillain-Barre Syndrome | |
| | CCI |
| Myasthenic Syndrome | |
| | CCI |
| Vasculitis | CCI |
| Meralikia | 001 |
| Myelitis | CCI |
| Meningitis | |
| | CCI |
| Rash | |
| CCI | |
| Pruritus | |
| Vitiligo | |
| Lichenoid keratosis | |
| Lichenoid Keratosis | CCI |
| Musculoskeletal pain | 301 |
| CCI | |
| Arthritis | CCI |
| Tendosynovitis | |
| | CCI |




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015): Kevnote-PN798 |
|---|---|---|---|
|---|---|---|---|

| irAEs (adverse reactions – at least possibly related to either pembro and/or efti) | |
|---|---|
| | Preferred Terms |
| Oedema | |
| CCI | |

#### **Notes:**

- Tables presented will contain both counts of subjects and events. Subjects who have multiple events in the same system organ class and preferred term will be counted only once in the subject counts.
- AEs coded using MedDRA version 21.1 or higher.
- Treatment-emergent principle All adverse events starting on or after first dosing are considered treatment-emergent adverse events (TEAE). All adverse events emerging during the screening period will only be listed, not presented in any of the tables. These events are no TEAEs. All tables will present TEAEs only.
- Treatment relatedness Following ICH-E3, the drug relatedness will be dichotomized as follows: Drug related: at least possibly drug related, OR with missing drug relatedness (= worst-case) Not drug related: not related. In tabulations this dichotomized parameter will be used, but in the listings the original parameter will be presented.
- Worst-case principle When cross-tabulating AE preferred terms versus an AE attribute (e.g., severity), the worst-case is always applied within each analysis period. I.e., when a subject has two times the same AE preferred term in the same analysis period, then the subject is reported only once: only with the worst severity. If this happens in two different analysis periods, the AE is reported twice; once in each analysis period. In the analysis the worst-case will be defined.

## 4.13.2 Laboratory Findings

Results (values and change from baseline) from the following laboratory parameters, recorded at screening and pre-dose on day 1 of each cycle except thyroid function tests which are performed at screening and every 2nd cycle starting with cycle 2, will be summarized by indication and visit.

#### Hematology:

Leukocytes/White blood cell (WBC) count with differential including absolute neutrophil count (ANC), absolute lymphocyte count, NLR ratio (absolute neutrophil count/ absolute lymphocyte count) absolute monocyte count, absolute eosinophil count, absolute basophil count; Erythrocytes/red blood cells (RBC) count, platelet count, hemoglobin and hematocrit.

#### **Biochemistry:**

Creatinine, random glucose, urea, alkaline phosphatase, alanine aminotransferase (ALT = GPT), aspartate aminotransferase (AST = GOT), gamma glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), total bilirubin, total protein, albumin/globulin ratio, sodium, potassium, chloride, calcium, phosphate, bicarbonates, uric acid, cholesterol, triglycerides, plasma amylase and c-reactive protein (CRP).

TPBS001 Version 6 (based on TPQA036 Version 2) CONFIDENTIAL



| Sponsor: | Immutep S.A.S. | I Protocol Killmaner. | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

Hepatic toxicity will be assessed based on the following Liver Function Tests (LFTs): Albumin, ALT, AST, ALP and Total Bilirubin (TBL). For these parameters, NCI-CTCAE grades are defined.

Tabulation of liver function parameters for Hy's law interpretations will be generated presenting frequencies of subjects with post-C1D1 parameters:

- Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) >3,
   >5, >10 and >20 times upper limit of the normal range (ULN), Bilirubin (BILI)
   >2x ULN;
- Simultaneous occurrence of ALT or AST >3x ULN and BILI >2.0x ULN;
- Simultaneous occurrence of ALT or AST >3x ULN and BILI >2.0x ULN subcategorized by ALP <2x ULN and >2x ULN.

Post-baseline potential Hy's Law cases will be identified using the following definition:

• either AST or ALT >  $3 \times ULN$  with concurrent ALP <  $2 \times ULN$  and concurrent total bilirubin  $\geq 2 \times ULN$ .

## Coagulation:

Prothrombin time (PT) and activated partial thromboplastin time (APTT).

## **Thyroid Function:**

Triiodothyronine (T3) or free triiodothyronine (FT3), free thyroxine (FT4) and thyroid stimulating hormone (TSH).

## **Urinalysis:**

Dipstick, *or* standard urinalysis (UA) with reflex microscopy and culture if clinically indicated. Gross urine examination (dipstick) and other tests should include visual inspection, pH, protein, ketones, glucose, bilirubin, nitrite, urobilinogen, occult blood, WBCs.

Changes from baseline will also be summarized where applicable.

Where applicable, CTCAE grades will be assigned to laboratory parameters. Certain parameters may have both high and low CTC grades assigned and where this occurs, high and low grades will be summarized separately. Shift tables comparing the worst post-baseline grade against the baseline grade will be prepared and will be provided for final analysis.

If possible, CTCAE Grade will be calculated for following parameters,

- Hematology parameters (all on two directions Low and High).
  - Leukocytes/White blood cell (WBC) count with differential including absolute neutrophil count (ANC), absolute lymphocyte count, ratio (absolute neutrophil count/ absolute lymphocyte count), absolute monocyte count, absolute eosinophil count, absolute basophil count; Erythrocytes/red blood cells (RBC) count, platelet count, hemoglobin and hematocrit.
- Biochemistry:
  - On two directions (Low and High): Creatinine, random glucose and urea;

TPBS001 Version 6 CONFIDENTIAL Effective Date: 15<sup>th</sup> March 2017 (based on TPQA036 Version 2) Prior Effective Date: 9<sup>th</sup> October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

On one direction (High): alkaline phosphatase, alanine aminotransferase (ALT = GPT), aspartate aminotransferase (AST = GOT), triglycerides and plasma amylase.

- Thyroid Function (all on two directions Low and High): Triiodothyronine (T3) or free triiodothyronine (FT3), free thyroxine (FT4) and thyroid stimulating hormone (TSH).

Categorical laboratory parameters will be summarized by shift tables comparing the result/abnormality at each visit against the result/abnormality at baseline.

Serology results at Screening are described in Section 4.4.

Pregnancy test results will be listed only.

#### **Notes:**

- All results outside predefined normal ranges will be flagged in the data listings;
- Repeat laboratory results within a visit will not be used in any summary calculations; Unscheduled and repeat results will be listed only;
- Any other laboratory results will be listed only;
- CTCAE Grade version 4.03 will be used for derivation of the laboratory parameters;

### 4.13.3 Vital Signs

Results for systolic and diastolic blood pressure, temperature, pulse rate, body weight and derived BMI will be summarized by indication and visit. Changes from baseline will also be summarized.

#### 4.13.4 ECG Results

The quantitative ECG assessments (heart rate, PR interval, RR interval, QRS duration and QT interval) will be summarized by indication and visit. Changes from baseline will also be summarized.

Investigator interpretation is collected for each parameter individually will be derived to create an overall investigator interpretation at each visit as,

- in case any of the parameters for the given ECG assessment is marked as "abnormal, clinically significant", the whole test should be considered as "abnormal, clinically significant";
- if none of the parameters are "abnormal, clinically significant" but at least one is indicated as "abnormal, not clinically significant", the whole ECG assessment should be considered as "abnormal, not clinically significant";
- if all the parameters are "normal", then the whole ECG assessment should be considered "normal";

The overall investigator interpretation will be listed.

#### 4.13.5 ECOG Performance Status

The number and percentage of subjects with each ECOG PS response at each visit will be presented. In addition, the number and percentage of subjects who have improved, deteriorated and stayed the same compared to baseline will be presented at each post-baseline visit.


Prior Effective Date: 9th October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321- |
|-----------|-------------------|-------------------|----------------------|
| Sporisor. | IIIIIIutep S.A.S. | FIOLOCOLINALIDEL. | P015); Keynote-PN798 |

## 4.13.6 Physical Examination

Data collected from the physical examination will be listed only.

## 4.14 Adjustment for Covariates

There is no statistical analysis planned and hence no adjustment for covariates.

#### 4.14.1 Center Effects

This study will be conducted at approximately 12 centers. Subjects from all centers will be pooled. No adjustment for centers will be conducted.

#### 4.15 Protocol Violations or Deviations

A protocol deviation (PD) list is created at beginning of the study to collect all PD identified on site and/data issue. The PD list is reviewed on an ongoing basis by sponsor and Fortrea team. During this review, the deviations are classified as important and non-important.

Important deviations will be tabulated and listed.

# 4.16 Handling of Missing Data

When tumor response (as defined by local image interpretation) based on target lesions is missing, it will be set to PD if the last non-missing observation is PD. No imputation will be used to manage any other patterns of missing data for tumor response (i.e., it will be censored in the efficacy analysis).

Partial dates will be imputed only to allow classification of medications as prior, used at study entry, concomitant or post-treatment and AEs as treatment-emergent or not. The following rules will apply:

## Medications:

- Start Dates:
  - Missing day will be imputed by 1<sup>st</sup> day of the month; if same month and year than the date of first dose then the date of first dose will be used.
  - Missing month will be imputed by January; if same year as first dose, then the date the date of first dose will be used.
  - For completely missing date, then date of first dose will be used.

#### o End Dates:

- Missing day will be imputed by last day of the month; if same month and year than date of the last intake of study drug then the date of last dose will be used.
- Missing month will be imputed by last month of the year; if same year as date of the last intake of study drug, then the date of last dose will be used.
- For completely missing date then no substitution (i.e., treatment considered as still ongoing)

If (partially) missing dates do not allow to allocate the therapy as the last prior to inclusion, then the therapy is assumed before therapy with non-missing date information. Therapy 30 days before last therapy record prior to inclusion (date of date of first dose) is also considered




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

as last therapy. In case there is more than one therapy with the same end date all are considered as last therapy prior to inclusion. For best overall response assessment recorded on the last therapy record prior to inclusion, only prior anticancer systemic regimens will be considered.

After the imputation of missing partial start date by date of first intake, if the start date is after the end date of medication, then the start data = end date;

#### • AEs:

• When AE start date time is missing, the AE will be allocated to the first treatment period in the study.

#### Start Dates:

- missing day will be imputed by 1<sup>st</sup> day of the month; if same month and year than the date of first dose then the date of first dose will be used.
- missing month will be imputed by January; if same year as first dose, then the date the date of first dose will be used.
- if date is completely missing the date of first dose will be used.
- This approach will ensure that AEs with partial dates are assigned as treatmentemergent if the partial date is ambiguous.

#### o End Dates:

- missing day will be imputed by last day of the month; If same month and year than last visit date, then last visit date will be used;
- missing month will be imputed by December; if same year than last visit date then the date last visit will be used.
- if date is completely missing the date of last visit will be used.
- Missing time will not be imputed.
- o Date of last visit is the date of last visit as recorded in eCRF.

Imputed dates will not be listed and will not be used to calculate any durations.

### 4.17 Deviations from SAP

Any deviations from the original statistical plan will be described and justified in the final CSR.

## 4.18 Changes in Conduct or Planned Analyzes from the Protocol

## 4.18.1 Confirmatory Pre-Baseline RECIST 1.1

A note to file was created to correct the following inconsistency in the eCRF.

On form "Confirmatory Pre-Baseline RECIST 1.1 Response Assessment" (form only applicable for Part B subjects) the following issues were noticed:

- 1. the lower header of the form "Confirmatory Pre-Baseline RECIST 1.1 Response Assessment" includes a typo "iRECIST 1.1" instead of "RECIST 1.1"
- 2. for target and non-target lesion evaluation the options in the drop-down menus are given as per iRECIST and not as per RECIST 1.1




| Sponsor: Immutep | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|
|---|---|---|

Both issues could only be solved with an eCRF update and migration, but sponsor confirmed that they do not want a migration to solve that issues at this time. The following solutions have been discussed and agreed:

Issue #1: The typo in the header can be accepted without any changes.

Issue #2: The inconsistent drop-down menus will remain as they are, and Statistics will hard code the information as following:

| Folder: Confirmatory Pre-Baseline Radiological Assessments Form: Confirmatory Pre-Baseline RECIST 1.1 Form header: CONFIRMATORY PRE-BASELINE iRECIST 1.1 RESPONSE ASSESSMENT Item: Evaluation of Target Lesions [CCPIR.CONFEVLTL] | |
|---|---|
| eCRF drop down menu options: | to be hard coded to: |
| (iCR) COMPLETE RESPONSE | (CR) COMPLETE RESPONSE |
| (iPR) PARTIAL RESPONSE | (PR) PARTIAL RESPONSE |
| (iUPD) UNCONFIRMED PROGRESSIVE DISEASE | (PD) PROGRESSIVE<br>DISEASE |
| (iCPD) CONFIRMED PROGRESSIVE DISEASE | (PD) PROGRESSIVE<br>DISEASE |
| (iSD) STABLE DISEASE | (SD) STABLE DISEASE |
| (NE) NOT EVALUABLE | (NE) NOT EVALUABLE |
| iNON-CR/iNON-PD | NON-CR/iNON-PD |

| Folder: Confirmatory Pre-Baseline Radiological Assessments Form: Confirmatory Pre-Baseline RECIST 1.1 Form header: CONFIRMATORY PRE-BASELINE iRECIST 1.1 RESPONSE ASSESSMENT Item: Evaluation of Non-Target Lesions [CCPIR.CONFEVLNTL] | |
|---|---|
| eCRF drop down menu options: | to be hard coded to: |
| (iCR) COMPLETE RESPONSE | (CR) COMPLETE RESPONSE |
| iNON-CR/iNON-PD | NON-CR/NON-PD |
| (iUPD) UNCONFIRMED PROGRESSIVE DISEASE | (PD) PROGRESSIVE<br>DISEASE |
| (iCPD) CONFIRMED PROGRESSIVE DISEASE | (PD) PROGRESSIVE<br>DISEASE |
| (NE) NOT EVALUABLE | (NE) NOT EVALUABLE |

#### 4.18.2 Per Protocol Analysis

The analysis for efficacy endpoints will not be repeated for per-protocol analysis population. Another population of analysis was derived, the Evaluable Analysis Set (EAS) is a subset of the FAS and includes all subjects who received at least one dose of trial drug and has at least one evaluable post-baseline tumor assessment. The analysis initially planned to be run in per protocol population will be run on the EAS, e.g. for ORR, DCR, TTR, DoR, PFS and OS.

TPBS001 Version 6 CONFIDENTIAL Effective Date: 15<sup>th</sup> March 2017 (based on TPQA036 Version 2) Prior Effective Date: 9<sup>th</sup> October 2016



| Sponsor: |
|----------|
|----------|

## 4.18.3 Non-CR/Non-PD in BICR

For BICR data patients with BOR of "Non-CR/Non-PD" are included in stable disease category, so, considered as part of the Disease Control Rate for both RECIST 1.1 and iRECIST Guidelines.

## 4.19 Algorithms/SAS Codes

• Tables that need descriptive statistics – continuous variables:

```
PROC UNIVARIATE DATA=dset NOPRINT;

VAR var1 var2 var3 ...varn;

BY byvar; (optional)

OUTPUT OUT=outname

N=n MEAN=mean MIN=min MAX=max MEDIAN=median STD=std;

RUN;

PROC UNIVARIATE DATA=dset NOPRINT;

VAR var1 var2 var3 ...varn;

BY byvar; (optional)

OUTPUT OUT=outname

N=n MEAN=mean MIN=min MAX=max MEDIAN=median STD=std

PPD

RUN:
```

Tables that need frequency counts:

```
PROC FREQ DATA=dset NOPRINT;
BY byvar; (optional)
TABLES var1*var2;
OUTPUT OUT=outname;
RUN;
```

• Tables that need exact or asymptotic 95% CIs between groups for proportions:

```
PROC FREQ DATA=dset;
BY byvar; (optional)
TABLES var1 * var2 / MEASURES RISKDIFF ALPHA= CCI
EXACT MEASURES;
RUN;
```

**Notes:** 1 Estimates are computed for 2x2 tables only

2 This code also gives exact 95% CIs within group for binomial proportions

• Tables that need 95% CIs within group for binomial proportions:

```
PROC FREQ DATA=dset;
BY byvar; (optional)
TABLES var1;
EXACT BINOMIAL;
RUN;
```

 Tables that need number of events/censored and probabilities of failure/survival at cut off times:

TPBS001 Version 6 CONFIDENTIAL Effective Date: 15<sup>th</sup> March 2017 (based on TPQA036 Version 2) Prior Effective Date: 9<sup>th</sup> October 2016



```
PROC LIFETEST DATA=dset OUTSURV=LIFE METHOD=LT INTERVALS=3,6,9,12, 18,24,;

TIME duration*censor (0 or 1);

ID subject;

STRATA treatment;
RUN;
```

• Tables that need life table with estimates of survival, with CIs and log rank test:

```
PROC LIFETEST DATA=dset OUTSURV=LIFE METHOD=KM;
TIME duration*censor (0 or 1);
ID subject;
STRATA treatment;
RUN;
```

• The geometric mean is the antilog of the arithmetic mean of the logs:

```
DATA dset;

SET dset old;

LOGx = LOG(x);

RUN;

PROC UNIVARIATE DATA=dset NOPRINT;

VAR LOGx;

OUTPUT OUT=outname

MEAN=logmean;

RUN;

DATA outname;

SET outname;

geomean = EXP(logmean);

RUN;
```



# 5 Tables and Listings

## 5.1 Table Format

All output will be produced using SAS version 9.4 or a later version.

In the top left portion of each table/listing, a *table/listing number* followed by the *title* of the table/listing will be presented. After the title line, optional *sub-title* or *population* information can be presented. Horizontal lines will appear before and after the column heading of the table/listing. *Footnotes* will be put under the main body of text at the bottom of the page.

The *sponsor name*, *protocol number*, programmers User ID, status of the table/listing (i.e., draft or final) and *SAS program name* will appear bottom left in a string and the *page number* will appear on the bottom right corner of each table/listing. The *date and time of creation* of table/listing will appear bottom left under the Sponsor name. The source listing number will appear in the bottom left.

A *landscape layout* is proposed for both table and listing presentations.

The *left* and *right margins* of all tables and listings will be a minimum of 2.1 cm from the left and 1.9cm from the right. The *top and bottom margins* will be a minimum 2.92cm. *Header and footer* will be both 1.27 cm.

There is no special requirement of *font type* and *size*, but an *8-point* font size for tables and *7-* or *8-point* for listings is proposed using *Courier New* font. A maximum SAS line size=141 and page size=44 for *8-point* font size, and line size=161 and page size=50 for *7-point* will be used to fit on both UK and US paper sizes.

In a listing, in the case that a subject's record has been continued to the next page, an appropriate identification (e.g., the subject ID number) must be presented at the beginning of that page.

## 5.2 Conventions

Unless otherwise specified, in summary tables of continuous variables, the minimum and maximum values will be displayed to the same number of decimal places as the raw data, the mean median and quartiles will be presented to one extra decimal place compared to the raw data, and the standard deviation will be displayed to two extra decimal places compared to the raw data. Wherever possible, data will be decimally aligned.

Unless otherwise specified frequency tabulations will be presented by number and percentage, where the percentage is presented in brackets to 1 decimal place.

P-values, if applicable, will be presented to 3 decimal places. If a p-value is less than 0.05 but is greater than or equal to 0.01, then an asterisk (\*) will be added next to this value. If a p-value is less than 0.01 but is greater than or equal to 0.001, then two asterisks (\*\*) will be added next to this value. Finally, if the p-value is less than 0.001 then three asterisks (\*\*\*) will be added next to this value and it will be presented as <0.001. If the rounded result is a value of 1.000, it will be displayed as >0.999. Any date information in the listing will use the *date9*. format, for example, 07MAY2002. In the listing, a unit associated with a variable will be presented only once within parentheses either below or next to that variable in the heading portion. If a parameter has multiple units, each unit will be displayed only once, as applicable.


CONFIDENTIAL Effective Date: 15<sup>th</sup> March 2017

Prior Effective Date: 9th October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

All tables will have their source listing referenced in a footnote. Listings should be sorted as described in the programming notes in the shells. For data collected over several visits, SDTM. VISITNUM should be used to sort by visit. All listings should have the source dataset (ADaM or SDTM) referenced in a footnote. All tables, listings and figures will be collated into Microsoft Word documents (tables and listings as per ICH E3 Structure and content of clinical study reports sections, one for figures).

#### 5.3 Tables

| Output Number | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.1.1.1 | Subject Disposition (All Subjects) | U | FU1 | |
| Table 14.1.1.2 | Subject Disposition by Country (All Subjects) | U | FU1 | |
| Table 14.1.1.3 | Subject Disposition by Center (All Subjects) | R | FU1 | |
| Table 14.1.1.4 | Important Protocol Violations (All Subjects) | U | FU1 | |
| Table 14.1.2.1.1 | Demographics and Baseline<br>Characteristics (Full Analysis Set) | U | FU1 | |
| Table 14.1.2.1.2 | Demographics and Baseline<br>Characteristics by PD-L1 (Central<br>results)— Part A Only | U | FU1 | |
| Table 14.1.2.1.3 | Demographics and Baseline<br>Characteristics by PD-L1 (Central or<br>Local results) – Part A Only (Full<br>Analysis Set) | R | FU1 | |
| Table 14.1.3.1 | Past Medical History (Full Analysis Set) | U | FU1 | |
| Table 14.1.3.2 | Concomitant Diseases (Full Analysis Set) | U | FU1 | |
| Table 14.1.4.1 | Cancer History (Full Analysis Set) | U | FU1 | |
| Table 14.1.4.2 | History of HIV, HCV, HBV (Full<br>Analysis Set) | U | FU1 | |
| Table 14.1.4.3 | Active Disease sites at Baseline (Full Analysis Set) | U | FU1 | |
| Table 14.1.5.1 | Previous Cancer Surgery, Radiotherapy<br>and Systemic Anti-cancer Therapy (Full<br>Analysis Set) | U | FU1 | |
| Table 14.1.5.2 | Previous systemic anti-cancer therapy (Full Analysis Set) | U | FU1 | |
| Table 14.1.6.1 | Prior Medications other than anti-cancer therapy (Full Analysis Set) | U | FU1 | |
| Table 14.1.6.2 | Medications used at study entry and<br>Concomitant Medications (Full<br>Analysis Set) | U | FU1 | |
| Table 14.1.7 | Concomitant Procedures (Full Analysis Set) | U | FU1 | |
| Table 14.1.8.1 | New Anti-cancer Therapy (Full<br>Analysis Set) | U | FU1 | |
| Table 14.1.8.2 | Subsequent anti-cancer procedures (Full Analysis Set) | U | FU1 | |




| Output Number | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.1.9.1 | Efti Exposure and Compliance (Full Analysis Set) | U | FU1 | |
| Table 14.1.9.2 | Pembrolizumab Exposure and<br>Compliance (Full Analysis Set) | U | FU1 | |
| Table 14.1.9.3 | Efti and Pembrolizumab Exposure and Compliance (Full Analysis Set) | R | FU1 | |
| Table 14.1.10.1 | Other Derived Variables (Full Analysis Set) | U | FU1 | |
| Table 14.2.1.1.1 | Overall Response Rate - iRECIST confirmed (Full Analysis Set) | U | FU1 | Yes |
| Table 14.2.1.1.2 | Overall Response Rate - iRECIST unconfirmed (Full Analysis Set) | R | FU1 | Yes |
| Table 14.2.1.1.3 | Overall Response Rate - RECIST 1.1 confirmed (Full Analysis Set) | R | FU1 | Yes |
| Table 14.2.1.1.4 | Overall Response Rate - RECIST 1.1 unconfirmed (Full Analysis Set) | R | FU1 | Yes |
| Table 14.2.1.2.1 | Overall Response Rate - iRECIST confirmed (Evaluable Analysis Set) | R | FU1 | Yes |
| Table 14.2.1.2.2 | Overall Response Rate - iRECIST unconfirmed (Evaluable Analysis Set) | R | FU1 | Yes |
| Table 14.2.1.2.3 | Overall Response Rate - RECIST 1.1 confirmed (Evaluable Analysis Set) | R | FU1 | Yes |
| Table 14.2.1.2.4 | Overall Response Rate - RECIST 1.1 unconfirmed (Evaluable Analysis Set) | R | FU1 | Yes |
| Table 14.2.2.1.1 | Duration of Response according to iRECIST (Full Analysis Set Responders Only) | U | FU1 | Yes |
| Table 14.2.2.1.2 | Duration of Response according to<br>RECIST 1.1 (Full Analysis Set -<br>Responders Only) | R | FU1 | Yes |
| Table 14.2.3.1.1 | Time to Response according to iRECIST (Full Analysis Set) | U | FU1 | Yes |
| Table 14.2.3.1.2 | Time to Response according to RECIST 1.1 (Full Analysis Set) | R | FU1 | Yes |
| Table 14.2.4.1.1 | Progression Free Survival according to iRECIST (Full Analysis Set) | U | FU1 | Yes |
| Table 14.2.4.1.2 | Progression Free Survival according to RECIST 1.1 (Full Analysis Set) | R | FU1 | Yes |
| Table 14.2.4.2.1 | Progression Free Survival according to iRECIST (Evaluable Analysis Set) | R | FU1 | Yes |
| Table 14.2.4.2.2 | Progression Free Survival according to RECIST 1.1 (Evaluable Analysis Set) | R | FU1 | Yes |
| Table 14.2.5.1 | Overall Survival (Full Analysis Set) | R | FU1 | |
| Table 14.2.6.1 | Autoantibodies and Anti-drug<br>Antibodies against Efti (Full Analysis<br>Set) | U | FU1 | |
| Table 14.2.7.1.1 | Circulating Biomarkers – Absolute<br>values and change from Baseline (Full<br>Analysis Set) | R | FU1 | |
| Table 14.2.7.1.2 | Circulating Biomarkers – Percentage change from Baseline (Full Analysis Set) | R | FU1 | |




| Output Number | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.2.8.1.1.1.1 | Overall Response Rate by PD-L1 –<br>Central - Part A: NSCLC 1st line (Full<br>Analysis Set) | U | FU1 | |
| Table 14.2.8.1.1.1.2 | Overall Response Rate by PD-L1 –<br>Central - Part C: HNSCC (Full Analysis<br>Set) | R | FU1 | |
| Table 14.2.8.1.1.2.1 | Overall Response Rate by PD-L1 -<br>Central or Local - Part A: NSCLC 1st<br>line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.1.2.2 | Overall Response Rate by PD-L1-<br>Central or Local- Part B: NSCLC 2nd<br>line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.2.1 | Overall Response Rate by Sex - Part A:<br>NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.2.2 | Overall Response Rate by Sex - Part B:<br>NSCLC 2nd line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.2.3 | Overall Response Rate by Sex - Part C:<br>HNSCC (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.3.1 | Overall Response Rate by Smoking<br>Status - Part A: NSCLC 1st line (Full<br>Analysis Set) | U | FU1 | |
| Table 14.2.8.1.3.2 | Overall Response Rate by Smoking<br>Status - Part B: NSCLC 2nd line (Full<br>Analysis Set) | R | FU1 | |
| Table 14.2.8.1.3.3 | Overall Response Rate by Smoking<br>Status - Part C: HNSCC (Full Analysis<br>Set) | R | FU1 | |
| Table 14.2.8.1.4.1 | Overall Response Rate by Age - Part A:<br>NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.4.2 | Overall Response Rate by Age - Part B:<br>NSCLC 2nd line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.4.3 | Overall Response Rate by Age - Part C:<br>HNSCC (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.5.1 | Overall Response Rate by ECOG Performance Status - Part A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.5.2 | Overall Response Rate by ECOG Performance Status - Part B: NSCLC 2nd line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.5.3 | Overall Response Rate by ECOG<br>Performance Status - Part C: HNSCC<br>(Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.6.1 | Overall Response Rate by Overall ADA - Part A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.6.2 | Overall Response Rate by Overall ADA - Part B: NSCLC 2nd line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.6.3 | Overall Response Rate by Overall ADA<br>- Part C: HNSCC (Full Analysis Set) | R | FU1 | |




| <b>Output Number</b> | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.2.8.1.7.1 | Overall Response Rate by Region - Part<br>A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.7.2 | Overall Response Rate by Region - Part<br>B: NSCLC 2nd line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.7.3 | Overall Response Rate by Region - Part<br>C: HNSCC (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.1.8.1 | Overall Response Rate by Tumor Type - Part A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.9.1 | Overall Response Rate by Resistance -<br>Part B: NSCLC 2nd line (Full Analysis<br>Set) | R | FU1 | |
| Table 14.2.8.1.10.1 | Overall Response Rate by Prior cetuximab - Part C: HNSCC (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.11.1 | Overall Response Rate by HPV status -<br>Part C: HNSCC (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.1.12.1 | Overall Response Rate by Prior<br>Therapy - Part B: NSCLC 2nd line (Full<br>Analysis Set) | U | FU1 | |
| Table 14.2.8.1.13.1 | Overall Response Rate by Maximum<br>Absolute Lymphocyte count (ALC)<br>change - Part A: NSCLC 1st line (Full<br>Analysis Set) | U | FU1 | |
| Table 14.2.8.1.13.2 | Overall Response Rate by Maximum<br>Absolute Lymphocyte count (ALC)<br>change - Part B: NSCLC 2nd line (Full<br>Analysis Set) | R | FU1 | |
| Table 14.2.8.1.13.3 | Overall Response Rate by Maximum<br>Absolute Lymphocyte count (ALC)<br>change - Part C: HNSCC (Full Analysis<br>Set) | R | FU1 | |
| Table 14.2.8.2.1.1.1 | Survival Analysis Endpoints by PD-L1 - Central - Part A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.1.1.2 | Survival Analysis Endpoints by PD-L1 – Central - Part C: HNSCC (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.1.2.1 | Survival Analysis Endpoints by PD-L1 — Central or Local - Part A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.1.2.2 | Survival Analysis Endpoints by PD-L1-<br>Central or Local- Part B: NSCLC 2nd<br>line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.2.1 | Survival Analysis Endpoints by Sex -<br>Part A: NSCLC 1st line (Full Analysis<br>Set) | U | FU1 | |
| Table 14.2.8.2.2.2 | Survival Analysis Endpoints by Sex -<br>Part B: NSCLC 2nd line (Full Analysis<br>Set) | R | FU1 | |
| Table 14.2.8.2.2.3 | Survival Analysis Endpoints by Sex -<br>Part C: HNSCC (Full Analysis Set) | R | FU1 | |




| Output Number | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.2.8.2.3.1 | Survival Analysis Endpoints by<br>Smoking Status - Part A: NSCLC 1st<br>line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.3.2 | Survival Analysis Endpoints by<br>Smoking Status - Part B: NSCLC 2nd<br>line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.3.3 | Survival Analysis Endpoints by<br>Smoking Status - Part C: HNSCC (Full<br>Analysis Set) | R | FU1 | |
| Table 14.2.8.2.4.1 | Survival Analysis Endpoints by Age -<br>Part A: NSCLC 1st line (Full Analysis<br>Set) | U | FU1 | |
| Table 14.2.8.2.4.2 | Survival Analysis Endpoints by Age -<br>Part B: NSCLC 2nd line (Full Analysis<br>Set) | R | FU1 | |
| Table 14.2.8.2.4.3 | Survival Analysis Endpoints by Age -<br>Part C: HNSCC (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.5.1 | Survival Analysis Endpoints by ECOG<br>Performance Status - Part A: NSCLC<br>1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.5.2 | Survival Analysis Endpoints by ECOG<br>Performance Status - Part B: NSCLC<br>2nd line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.5.3 | Survival Analysis Endpoints by ECOG<br>Performance Status - Part C: HNSCC<br>(Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.6.1 | Survival Analysis Endpoints by Overall<br>ADA - Part A: NSCLC 1st line (Full<br>Analysis Set) | U | FU1 | |
| Table 14.2.8.2.6.2 | Survival Analysis Endpoints by Overall<br>ADA - Part B: NSCLC 2nd line (Full<br>Analysis Set) | R | FU1 | |
| Table 14.2.8.2.6.3 | Survival Analysis Endpoints by Overall<br>ADA - Part C: HNSCC (Full Analysis<br>Set) | R | FU1 | |
| Table 14.2.8.2.7.1 | Survival Analysis Endpoints by Region - Part A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.7.2 | Survival Analysis Endpoints by Region - Part B: NSCLC 2nd line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.7.3 | Survival Analysis Endpoints by Region - Part C: HNSCC (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.8.1 | Survival Analysis Endpoints by Tumor<br>Type - Part A: NSCLC 1st line (Full<br>Analysis Set) | U | FU1 | |
| Table 14.2.8.2.9.1 | Survival Analysis Endpoints by<br>Resistance - Part B: NSCLC 2nd line<br>(Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.10.1 | Survival Analysis Endpoints by Prior<br>cetuximab - Part C: HNSCC (Full<br>Analysis Set) | U | FU1 | |




| Output Number | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.2.8.2.11.1 | Survival Analysis Endpoints by HPV status - Part C: HNSCC (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.12.1 | Survival Analysis Endpoints by Prior<br>Therapy - Part B: NSCLC 2nd line (Full<br>Analysis Set) | U | FU1 | |
| Table 14.2.8.2.13.1 | Survival Analysis Endpoints by Maximum Absolute Lymphocyte count (ALC) change - Part A: NSCLC 1st line (Full Analysis Set) | U | FU1 | |
| Table 14.2.8.2.13.2 | Survival Analysis Endpoints by<br>Maximum Absolute Lymphocyte count<br>(ALC) change - Part B: NSCLC 2nd<br>line (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.2.13.3 | Survival Analysis Endpoints by Maximum Absolute Lymphocyte count (ALC) change - Part C: HNSCC (Full Analysis Set) | R | FU1 | |
| Table 14.2.8.3.1 | Overall Survival (OS) by Response -<br>Part A: NSCLC 1st line (Full Analysis<br>Set) | U | FU1 | |
| Table 14.2.8.3.2 | Overall Survival (OS) by Response -<br>Part B: NSCLC 2nd line (Full Analysis<br>Set) | U | FU1 | |
| Table 14.2.8.3.3 | Overall Survival (OS) by Response -<br>Part C: HNSCC (Full Analysis Set) | U | FU1 | |
| Table 14.2.9.1.1 | CCI | R | FU1 | |
| Table 14.3.1.1 | Summary of Treatment-emergent Adverse Events (Safety Population) | U | FU1 | |
| Table 14.3.1.2 | Treatment-emergent Adverse Events by<br>System Organ Class and Preferred Term<br>(Safety Population) | U | FU1 | |
| Table 14.3.1.3 | Tabulation of all treatment-related Treatment-emergent adverse events (Safety Population) | U | FU1 | |
| Table 14.3.1.4 | Serious Treatment-emergent Adverse<br>Events by System Organ Class and<br>Preferred Term (Safety Population) | R | FU1 | |
| Table 14.3.1.5 | Fatal Treatment-emergent Adverse<br>Events by System Organ Class and<br>Preferred Term (Safety Population) | R | FU1 | |
| Table 14.3.1.6 | Treatment-emergent Adverse Events Leading to Permanent Discontinuation of Efti by System Organ Class and Preferred Term (Safety Population) | R | FU1 | |
| Table 14.3.1.7 | Treatment-emergent Adverse Events Leading to Permanent Discontinuation of Pembrolizumab by System Organ Class and Preferred (Safety Population) | R | FU1 | |


Prior Effective Date: 9th October 2016



| Output Number | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.3.1.8 | Treatment-emergent Adverse Events<br>Leading to Discontinuation from Study<br>by System Organ Class and Preferred<br>Term (Safety Population) | R | FU1 | |
| Table 14.3.1.9 | Treatment-emergent Events of Clinical<br>Interest by System Organ Class and<br>Preferred Term (Safety Population) | R | FU1 | |
| Table 14.3.1.10 | Treatment-emergent Adverse Events by<br>Severity, System Organ Class and<br>Preferred Term (Safety Population) | U | FU1 | |
| Table 14.3.1.11 | Local injection site reactions Treatment-<br>emergent Adverse Events by Severity,<br>System Organ Class and Preferred Term<br>(Safety Population) | R | FU1 | |
| Table 14.3.1.12 | Treatment-emergent Adverse Events irrespective of relatedness to study drug by Severity, System Class and Preferred Term (Safety Population) | R | FU1 | |
| Table 14.3.1.13 | Treatment-emergent Adverse Events related to Eftilagimod and/or Pembrolizumab by Severity, System Class and Preferred Term (Safety Population) | R | FU1 | |
| Table 14.3.1.14 | Treatment-emergent systemic inflammatory response events with in 24 hrs from efti administration (Safety Population) | R | FU1 | |
| Table 14.3.1.15 | Treatment-emergent irAEs (Adverse reactions – Related to either pembro and/or efti) (Safety Population) | R | FU1 | |
| Table 14.3.1.16 | Treatment Emergent Adverse events with CTCAE Grade ≥ 3 by system organ class and preferred term (Safety Population) | R | FU1 | |
| Table 14.3.1.17 | Treatment Emergent Adverse events with CTCAE Grade ≥ 3 by Relationship to Efti, to pembro, to efti and/or pembro by System Organ Class and Preferred Term (Safety Population) | R | FU1 | |
| Table 14.3.5.1.1 | Hematology Results and Changes from Baseline (Safety Population) | U | FU1 | |
| Table 14.3.5.1.2 | Biochemistry Results and Changes from Baseline (Safety Population) | R | FU1 | |
| Table 14.3.5.1.3 | Coagulation Results and Changes from Baseline (Safety Population) | R | FU1 | |
| Table 14.3.5.1.4 | Thyroid Function Results and Changes from Baseline (Safety Population) | R | FU1 | |
| Table 14.3.5.1.5 | Microscopic Urinalysis Results and<br>Changes from Baseline (Safety<br>Population) | R | FU1 | |
| Table 14.3.5.2 | Liver Function Test Elevations (Safety Population) | U | FU1 | |


Prior Effective Date: 9th October 2016



| Output Number | Output Title | U/R | Analysis | BICR data |
|---|---|---|---|---|
| Table 14.3.5.3.1 | Shift Table of Laboratory Test Results<br>between Baseline and worst NCI-<br>CTCAE grading – Hematology (Safety<br>Population) | U | FU1 | |
| Table 14.3.5.3.2.1 | Shift Table of Laboratory Test Results<br>between Baseline and worst NCI-<br>CTCAE grading – Biochemistry I<br>(Safety Population) | R | FU1 | |
| Table 14.3.5.3.2.2 | Shift Table of Laboratory Test Results<br>between Baseline and worst NCI-<br>CTCAE grading – Biochemistry II<br>(Safety Population) | U | FU1 | |
| Table 14.3.5.3.2.3 | Shift Table of Laboratory Test Results<br>between Baseline and worst NCI-<br>CTCAE grading – Thyroid Function<br>(Safety Population) | R | FU1 | |
| Table 14.3.5.3.3 | Laboratory Results – Hematology –<br>Shift Table (Safety Population) | U | FU1 | |
| Table 14.3.5.3.4 | Laboratory Results – Biochemistry –<br>Shift Table (Safety Population) | R | FU1 | |
| Table 14.3.5.3.5 | Laboratory Results – Coagulation –<br>Shift Table (Safety Population) | R | FU1 | |
| Table 14.3.5.3.6 | Laboratory Results – Thyroid Function – Shift Table (Safety Population) | R | FU1 | |
| Table 14.3.5.3.7 | Laboratory Results – Urinalysis – Shift Table (Safety Population) | R | FU1 | |
| Table 14.3.6 | Vital Signs Results and Changes from Baseline (Safety Population) e | U | FU1 | |
| Table 14.3.7 | 12-lead ECG Results and Changes from Baseline (Safety Population) | U | FU1 | |
| Table 14.3.8.1 | ECOG Performance Status (Safety Population) | U | FU1 | |

FU1 = Follow up analysis 1



# 5.4 Listings

| Output Number | Output Title | U/R | Analysis | BICR<br>data |
|---|---|---|---|---|
| Listing 14.3.2.1 | Listing of Deaths | U | FU1 | |
| Listing 14.3.2.2 | Listing of Fatal Treatment-emergent Adverse<br>Events | U | FU1 | |
| Listing 14.3.2.3 | Listing of Serious Treatment-emergent Adverse<br>Events | R | FU1 | |
| Listing 14.3.2.4.1 | Listing of Treatment-emergent Adverse Events Leading to Discontinuation from treatment (efti or Pembro) | R | FU1 | |
| Listing 14.3.2.4.2 | Listing of Treatment-emergent Adverse Events<br>Leading to Discontinuation from Study | U | FU1 | |
| Listing 14.3.2.5 | Listing of Treatment-emergent Events of Clinical Interest | R | FU1 | |
| Listing 14.3.4 | Listing of Abnormal Laboratory Results | U | FU1 | |
| Listing 16.2.1.1 | Subject Disposition | U | FU1 | |
| Listing 16.2.1.2 | Listing of subjects who permanently discontinued treatment Efti and Pembro (Safety Population) | R | FU1 | |
| Listing 16.2.2 | Important Protocol Deviations | U | FU1 | |
| Listing 16.2.3 | Exclusions from Analysis Populations | U | FU1 | |
| Listing 16.2.4.1 | Demographics/Baseline Characteristics | U | FU1 | |
| Listing 16.2.4.2 | Smoking History | U | FU1 | |
| Listing 16.2.4.3 | Medical/Surgical History | U | FU1 | |
| Listing 16.2.4.4.1 | Cancer History – Part I | U | FU1 | |
| Listing 16.2.4.4.2 | Cancer History – Part II | U | FU1 | |
| Listing 16.2.4.5 | History of HIV, HCV, HBV, HPV and PD-L1 | U | FU1 | |
| Listing 16.2.4.6 | Prior and Subsequent Cancer Surgery | U | FU1 | |
| Listing 16.2.4.7 | Prior Radiotherapy | U | FU1 | |
| Listing 16.2.4.8 | Prior Systemic Anti-cancer Therapy | U | FU1 | |
| Listing 16.2.4.9 | Medications | U | FU1 | |
| Listing 16.2.4.10 | Concomitant Surgical/Medical Procedures | U | FU1 | |
| Listing 16.2.4.11 | Other Derived Variables – Subgroup Variable | U | FU1 | |
| Listing 16.2.4.12 | Other Derived Variables – Subgroup Lab parameters | U | FU1 | |
| Listing 16.2.5.1 | Efti Administration, Exposure and Compliance | U | FU1 | |
| Listing 16.2.5.2 | Pembrolizumab Administration, Exposure and Compliance | U | FU1 | |
| Listing 16.2.5.3 | Visit Dates | U | FU1 | |
| Listing 16.2.5.4 | Comments | U | FU1 | |
| Listing 16.2.6.1 | Target Lesions | U | FU1 | Yes |
| Listing 16.2.6.2 | Non-target Lesions | U | FU1 | Yes |
| Listing 16.2.6.3 | New Lesions | U | FU1 | Yes |




| Output Number | Output Title | U/R | Analysis | BICR<br>data |
|---|---|---|---|---|
| Listing 16.2.6.4 | Assessment of Anti-Tumor Activity | U | FU1 | Yes |
| Listing 16.2.6.5 | Derived Efficacy Results | U | FU1 | Yes |
| Listing 16.2.6.6 | New Systemic Anti-cancer Therapy | U | FU1 | |
| Listing 16.2.6.7 | Immunogenicity Results (Autoantibodies and Anti-drug Antibodies against Efti) | U | FU1 | |
| Listing 16.2.6.8 | Circulating Biomarker Results | U | FU1 | |
| Listing 16.2.6.9 | Tumor Growth Kinetics | U | FU1 | Yes |
| Listing 16.2.6.10 | Subsequent anti-cancer procedures | U | | |
| Listing 16.2.7.1 | Adverse Events | R | FU1 | |
| Listing 16.2.7.2 | Listing of local injection site reactions | R | FU1 | |
| Listing 16.2.7.3 | Adverse events meeting the SMQ "Hypersensitivity" | R | FU1 | |
| Listing 16.2.7.4 | Systemic inflammatory response event with in 24 hrs from efti intake | U | FU1 | |
| Listing 16.2.7.5 | Treatment-emergent irAEs (Adverse reactions – Related to either pembro and/or efti) | R | FU1 | |
| Listing 16.2.8.1 | Laboratory Results - Hematology | U | FU1 | |
| Listing 16.2.8.2 | Laboratory Results – Biochemistry | R | FU1 | |
| Listing 16.2.8.3 | Laboratory Results – Thyroid Function | R | FU1 | |
| Listing 16.2.8.4 | Laboratory Results – Coagulation | R | FU1 | |
| Listing 16.2.8.5 | Laboratory Results - Urinalysis | U | FU1 | |
| Listing 16.2.8.6 | Pregnancy Test | U | FU1 | |
| Listing 16.2.8.7 | Vital Signs | U | FU1 | |
| Listing 16.2.8.8 | 12-lead ECG | U | FU1 | |
| Listing 16.2.8.9 | ECOG Performance Status | U | FU1 | |
| Listing 16.2.8.10 | Physical Examination | U | FU1 | |

FU1 = Follow up analysis 1



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

# 5.5 Figures

| Output Number | Output Title | U/R | Analysis | BICR<br>data |
|---|---|---|---|---|
| | Duration of Response according to iRECIST -<br>Investigator (Part A - Full Analysis Set - Responders | | | |
| Figure 14.2.1.1.1 | Only) Duration of Response according to iRECIST - | U | FU1 | |
| | Investigator (Part C - Full Analysis Set - Responders | | | |
| Figure 14.2.1.1.2 | Only) | R | FU1 | |
| | Duration of Response according to RECIST 1.1 - | | | |
| E' 140112 | Investigator (Part A - Full Analysis Set - Responders | D | TT 11 | |
| Figure 14.2.1.1.3 | Only) Duration of Response according to RECIST 1.1 - | R | FU1 | |
| | Investigator (Part C - Full Analysis Set - Responders | | | |
| Figure 14.2.1.1.4 | Only) | R | FU1 | |
| | Duration of Response according to iRECIST | | | |
| | (Investigator) by PD-L1 central (Part A) (Full | | | |
| Figure 14.2.1.2.1 | Analysis Set - Responders Only) | U | FU1 | |
| | Duration of Response according to RECIST 1.1 | | | |
| Eiguro 14 2 1 2 2 | (Investigator) by PD-L1 central (Part A) (Full | D | FU1 | |
| Figure 14.2.1.2.2 | Analysis Set - Responders Only) Duration of Response according to iRECIST | R | FUI | |
| | (Investigator) by PD-L1 central or local (Part A) (Full | | | |
| Figure 14.2.1.2.3 | Analysis Set - Responders Only) | R | FU1 | |
| | Duration of Response according to RECIST 1.1 | | | |
| | (Investigator) by PD-L1 central or local (Part A) (Full | | | |
| Figure 14.2.1.2.4 | Analysis Set - Responders Only) | R | FU1 | |
| | Duration of Response according to iRECIST | | | |
| E' 142125 | (Investigator) by PD-L1 central (Part C) (Full | D | T21 11 | |
| Figure 14.2.1.2.5 | Analysis Set - Responders Only) Duration of Response according to RECIST 1.1 | R | FU1 | |
| | (Investigator) by PD-L1 central (Part C) (Full | | | |
| Figure 14.2.1.2.6 | Analysis Set - Responders Only) | R | FU1 | |
| 8 | Progression Free Survival according to iRECIST - | | | |
| Figure 14.2.2.1.1 | Investigator (Part A - Full Analysis Set) | U | FU1 | |
| | Progression Free Survival according to iRECIST - | | | |
| Figure 14.2.2.1.2 | Investigator (Part B - Full Analysis Set) | R | FU1 | |
| | Progression Free Survival according to iRECIST - | | | |
| Figure 14.2.2.1.3 | Investigator (Part C - Full Analysis Set) | R | FU1 | |
| | Progression Free Survival according to RECIST 1.1 - | | | |
| Figure 14.2.2.1.4 | Investigator (Part A - Full Analysis Set) | R | FU1 | |
| G | Progression Free Survival according to RECIST 1.1 - | 1 | = = = | |
| Figure 14.2.2.1.5 | Investigator (Part B - Full Analysis Set) | R | FU1 | |
| G | Progression Free Survival according to RECIST 1.1 - | | = = = | |
| Figure 14.2.2.1.6 | Investigator (Part C - Full Analysis Set) | R | FU1 | |
| <i>G.</i> | Progression Free Survival according to iRECIST - | | | |
| Figure 14.2.2.2.1 | Investigator (Part A – Evaluable Analysis Set) | R | FU1 | |
| | Progression Free Survival according to iRECIST - | 1 | | |
| Figure 14.2.2.2.2 | Investigator (Part B - Evaluable Analysis Set) | R | FU1 | |
| TPBS001 Version 6 | CONFIDENTIAL | | ive Date: 15 <sup>th</sup> | Marah 2017 |




| Output Number | Output Title | U/R | Analysis | BICR<br>data |
|---|---|---|---|---|
| Figure 14.2.2.2.3 | Progression Free Survival according to iRECIST - Investigator (Part C - Evaluable Analysis Set) | R | FU1 | |
| Figure 14.2.2.2.4 | Progression Free Survival according to RECIST 1.1 - Investigator (Part A - Evaluable Analysis Set) | R | FU1 | |
| Figure 14.2.2.2.5 | Progression Free Survival according to RECIST 1.1 - Investigator (Part B - Evaluable Analysis Set) | R | FU1 | |
| Figure 14.2.2.2.6 | Progression Free Survival according to RECIST 1.1 - Investigator (Part C - Evaluable Analysis Set) Progression Free Survival according to iRECIST | R | FU1 | |
| Figure 14.2.2.3.1.1 | (Investigator) by PD-L1 central (Part A - Full Analysis Set) Progression Free Survival according to RECIST 1.1 | U | FU1 | |
| Figure 14.2.2.3.1.2 | (Investigator) by PD-L1 central (Part A - Full<br>Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.1.3 | Progression Free Survival according to iRECIST (Investigator) by PD-L1 central or local (Part A - Full Analysis Set) Progression Free Survival according to RECIST 1.1 | R | FU1 | |
| Figure 14.2.2.3.1.4 | (Investigator) by PD-L1 central or local (Part A - Full Analysis Set) Progression Free Survival according to iRECIST | R | FU1 | |
| Figure 14.2.2.3.1.5 | (Investigator) by Tumor type (Part A - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.1.6 | Progression Free Survival according to RECIST 1.1 (Investigator) by Tumor type (Part A - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.1.7 | Progression Free Survival according to iRECIST (Investigator) by ALC Change (Part A - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.1.8 | Progression Free Survival according to RECIST 1.1 (Investigator) by ALC Change (Part A - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.2.1 | Progression Free Survival according to iRECIST (Investigator) by PD-L1 central or local (Part B - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.2.2 | Progression Free Survival according to RECIST 1.1 (Investigator) by PD-L1 central or local (Part B - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.2.3 | Progression Free Survival according to iRECIST (Investigator) by tumor resistance (primary vs secondary) (Part B - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.2.4 | Progression Free Survival according to RECIST 1.1 (Investigator) by tumor resistance (primary vs secondary) (Part B - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.2.5 | Progression Free Survival according to iRECIST (Investigator) by Prior Therapy (Part B - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.2.6 | Progression Free Survival according to RECIST 1.1 (Investigator) by Prior Therapy (Part B - Full Analysis Set) | R | FU1 | |




| Output Number | Output Title | U/R | Analysis | BICR<br>data |
|---|---|---|---|---|
| Figure 14.2.2.3.2.7 | Progression Free Survival according to iRECIST (Investigator) by ALC Change (Part B - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.2.7 | Progression Free Survival according to RECIST 1.1 (Investigator) by ALC Change (Part B - Full Analysis | K | 101 | |
| Figure 14.2.2.3.2.8 | / | R | FU1 | |
| Figure 14.2.2.3.3.1 | Progression Free Survival according to iRECIST (Investigator) by PD-L1 central (Part C - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.3.2 | Progression Free Survival according to RECIST 1.1 (Investigator) by PD-L1 central (Part C - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.3.3 | Progression Free Survival according to iRECIST (Investigator) by Maximum ALC Change (Part C - Full Analysis Set) | R | FU1 | |
| Figure 14.2.2.3.3.4 | Progression Free Survival according to RECIST 1.1 (Investigator) by Maximum ALC Change (Part C - Full Analysis Set) | R | FU1 | |
| Figure 14.2.3.1.1 | Overall Survival Part A (Full Analysis Set) | U | FU1 | |
| Figure 14.2.3.1.2 | Overall Survival Part B (Full Analysis Set) | R | FU1 | |
| Figure 14.2.3.1.3 | Overall Survival Part C (Full Analysis Set) | R | FU1 | |
| Figure 14.2.3.2.1.1 | Overall Survival by PD-L1 central (Part A - Full Analysis Set) | U | FU1 | |
| Figure 14.2.3.2.1.2 | Overall Survival by PD-L1 central or local (Part A - Full Analysis Set) | R | FU1 | |
| Figure 14.2.3.2.1.3 | Overall Survival by Tumor type (Part A - Full Analysis Set) | R | FU1 | |
| Figure 14.2.3.2.1.4 | | R | FU1 | |
| Figure 14.2.3.2.2.1 | Overall Survival by PD-L1 central or local (Part B - Full Analysis Set) | R | FU1 | |
| Figure 14.2.3.2.2.2 | Overall Survival by tumor resistance (primary vs secondary) (Part B - Full Analysis Set) Overall survival by prior therapy (Part B – Full | R | FU1 | |
| Figure 14.2.3.2.2.3 | Analysis Set) | R | FU1 | |
| Figure 14.2.3.2.2.4 | <b>3</b> / | R | FU1 | |
| Figure 14.2.3.2.3.1 | Overall Survival by PD-L1 central only (Part C - Full Analysis Set) | R | FU1 | |
| Figure 14.2.3.2.3.2 | Overall Survival by ALC Change (Part C - Full | R | FU1 | |
| Figure 14.2.4.1 | according to RECIST 1.1 (Investigator) (Part A - Full Analysis Set) | U | FU1 | |
| Figure 14.2.4.2 | · · | R | FU1 | |
| Figure 14.2.4.3 | CCI according to RECIST 1.1 (Investigator) (Part C - Full Analysis Set) | R | FU1 | |




| Output Number | Output Title | U/R | Analysis | BICR<br>data |
|---|---|---|---|---|
| Figure 14.2.5.1 | Waterfall Plot of Best Percent Change from Baseline of Sum of Target Lesion Diameters (Investigator) by PD-L1 central or local - Part A (Full Analysis Set) | U | FU1 | |
| Figure 14.2.5.2 | Waterfall Plot of Best Percent Change from Baseline of Sum of Target Lesion Diameters (Investigator) by PD-L1 central or local - Part B (Full Analysis Set) | R | FU1 | |
| Figure 14.2.5.3 | Waterfall Plot of Best Percent Change from Baseline of Sum of Target Lesion Diameters (Investigator) by PD-L1 central or local - Part C (Full Analysis Set) | R | FU1 | |
| Figure 14.2.6.1 | Variation of sum of best target lesions (iRECIST)<br>(Investigator) Part B (Full Analysis Set) | U | FU1 | |
| Figure 14.2.6.2 | Variation of sum of best target lesions (iRECIST) (BICR) Part B (Full Analysis Set) Box Plot of ALC Change by confirmed iBOR | R | FU1 | Yes |
| Figure 14.2.7.1.1 | (iCR+iPR vs Others) - iRECIST - Part A (Full Analysis Set) Box Plot of ALC Change by confirmed Best Disease | U | FU1 | Yes |
| Figure 14.2.7.1.2 | Control (iCR+iPR+iSD vs Others) - iRECIST - Part<br>A | U | FU1 | Yes |
| Figure 14.2.7.2.1 | Box Plot of ALC Change by confirmed iBOR (iCR+iPR vs Others) - iRECIST - Part B (Full Analysis Set) | R | FU1 | Yes |
| Figure 14.2.7.2.2 | Box Plot of ALC Change by confirmed Best Disease<br>Control (iCR+iPR+iSD vs Others) - iRECIST - Part B<br>Box Plot of ALC Change by confirmed iBOR | R | FU1 | Yes |
| Figure 14.2.7.3.1 | (iCR+iPR vs Others) - iRECIST - Part C (Full Analysis Set) Box Plot of ALC Change by confirmed Best Disease | R | FU1 | Yes |
| Figure 14.2.7.3.2 | Control (iCR+iPR+iSD vs Others) - iRECIST - Part C<br>(Full Analysis Set) | R | FU1 | Yes |
| Figure 14.2.8.1.1 | Overall Survival Kaplan-Meier plot by iBOR (confirmed iCR+iPR vs Unconfirmed iPR+iSD vs iPD+iNA/NE) – Investigator – iRECIST - Part A (Full Analysis Set) | U | FU1 | |
| Figure 14.2.8.1.2 | Overall Survival Kaplan-Meier plot by iBOR (confirmed iPR+iSD vs iPD+iNA/NE) – Investigator – iRECIST - Part B (Full Analysis Set) | U | FU1 | |
| Figure 14.2.8.1.3 | Overall Survival Kaplan-Meier plot by iBOR (confirmed iCR+iPR vs Unconfirmed iPR+iSD+PD+NA/NE) – Investigator - iRECIST - Part C (Full Analysis Set) | U | FU1 | |

FU1 = Follow up analysis 1

Tables, Listings, and Figures will follow the format of:

- TACTI002\_(P015)\_Version\_3 \_Shells\_31Jan2024;




# 5.6 Appendices

# 5.6.1 Tumor growth kinetics analysis in Part B - List of patients and their lesions

List of patients and their lesions which should be part of Tumor growth kinetics analysis in Part B are indicated in bold font.

| Pt ID | Confirmatory Pre-baseline target lesions (reference scan) | Baseline target lesions | Comments |
|---|---|---|---|
| AU0111 | LIVER 4A | LIVER Seg 4A/VIII | LIVER 4A only |
| | LIVER Seg VII/VIII | LIVER Seg V | - |
| | OTHER Kidney RIGHT | LYMPH NODE Para- | - |
| | | aortic | |
| AU0204 | LUNG Left lower lobe lung nodule<br>LEFT | LUNG Subpleural nodule right lower lung lobe RIGHT | Yes but only these two: |
| | LYMPH NODE Anterior mediastinal lymph node | LUNG Left Lower lobe<br>nodule LEFT | LUNG Left lower lobe lung nodule LEFT LYMPH NODE Anterior mediastinal lymph node |
| | | LYMPH NODE Anterior mediastinal lymph node | |
| | | LYMPH NODE Retrocrural Lymph Node | |
| AU0208 | LUNG Right Lung Lower Lobe RIGHT | LUNG Right lower lobe<br>RIGHT | Yes, both lesions |
| | LUNG Left Lung Lower Lobe LEFT | LUNG Left lower lobe<br>LEFT | |
| ES1104 | N/A | LUNG left hilar lung<br>LEFT<br>LYMPH NODE left | No |
| | | supraclavicular lymph<br>node LEFT | |
| ES1117 | LUNG lower right lobe RIGHT | LYMPH NODE under the chin | Yes but only LUNG lower right |
| | LYMPH NODE right hilar RIGHT | LUNG lower right lobe<br>RIGHT | lobe RIGHT |
| | OTHER pleura RIGHT | LUNG post-costophrenic<br>in lower right lobe<br>RIGHT | |
| | SUPRARENAL GLAND right adrenal RIGHT | | |
| | SUPRARENAL GLAND left adrenal LEFT | | |
| ES1151 | LUNG upper right lobe RIGHT | LYMPH NODE left subcarinal LEFT | |

TPBS001 Version 6 CONFIDENTIAL (based on TPQA036 Version 2)

Prior Effective Date: 9th October 2016



| Pt ID | Confirmatory Pre-baseline target lesions (reference scan) | Baseline target lesions | Comments |
|---|---|---|---|
| | (************************************** | LUNG upper right lobe<br>RIGHT | Yes but only<br>LUNG upper right<br>lobe RIGHT |
| ES1319 | N/A | LYMPH NODE Hilium<br>RIGHT | No |
| ES1406 | LUNG left upper lobe mass LEFT | OTHER right laterocervical mass RIGHT LUNG left lower lobe mass LEFT CHEST WALL lower | No |
| ES1423 | CHEST WALL left hiliar mass LEFT | periesophagic mass CHEST WALL superior pleuropulmonar mass LEFT CHEST WALL pleuropulmonar caudal metastasis LEFT LIVER liver metastasis next to sickle ligament RIGHT OTHER kidney metastasis LEFT | No |
| ES1424 | LUNG left parahiliar lung mass LEFT | LUNG left parahiliar<br>lung mass LEFT | Yes but only<br>LUNG left |
| | LUNG right upper lobe mass RIGHT | LUNG right lower lobe lung mass RIGHT LIVER liver metastasis on S.VIII RIGHT LIVER liver metastasis on S.IV RIGHT OTHER umbilical implant NOT APPLICABLE | parahiliar lung<br>mass LEFT |
| ES1429 | N/A | LYMPH NODE left hiliar<br>lymph node LEFT<br>LYMPH NODE<br>subcarinal lymph node<br>LUNG right hiliar lung<br>mass RIGHT | No |
| ES1430 | LUNG right lower lobe lung mass RIGHT LYMPH NODE right hiliar lymph node RIGHT | LUNG right lower lobe<br>lung mass RIGHT<br>LYMPH NODE right<br>hiliar lymph node<br>RIGHT | Yes |
| ES1434 | LUNG lung mass RIGHT | LUNG lung mass RIGHT OTHER pancreatic area BONE right iliac mass with soft tissue RIGHT | Yes but only<br>LUNG lung mass<br>RIGHT |
| UK2106 | LYMPH NODE Precarinal lymph node | LUNG Left upper lobe<br>lung nodule LEFT | |




| Pt ID | Confirmatory Pre-baseline target lesions (reference scan) | Baseline target lesions | Comments |
|---|---|---|---|
| | LYMPH NODE Aortopulmonary lymph node | LYMPH NODE Anterior mediastinal, retrosternal, node | Yes, but only left<br>upper lobe lung<br>lesion |
| | LUNG Left upper lobe spiculated lung mass LEFT | LYMPH NODE Peripancreatic node | |
| | | OTHER Peritoneal nodule right flank RIGHT | |
| UK2107 | SUPRARENAL GLAND Right adrenal mass RIGHT | SUPRARENAL<br>GLAND Right adrenal<br>mass RIGHT | Yes |
| | SUPRARENAL GLAND Left adrenal mass LEFT | SUPRARENAL GLAND Left adrenal mass LEFT | |
| UK2108 | N/A | LYMPH NODE<br>Supraclavicular fossa<br>lymph node LEFT | No |
| UK2109 | LYMPH NODE Right lower paratracheal node RIGHT | LYMPH NODE Subcarinal node | No |
| | LYMPH NODE Right upper paratracheal node RIGHT | LYMPH NODE Right paratracheal node RIGHT | |
| | | LUNG Left lower lobe<br>lung metastasis LEFT | |
| UK2110 | LUNG Right upper lobe lung mass RIGHT | LUNG Upper Lobe<br>RIGHT | Yes |
| UK2116 | N/A | LUNG Right lower lobe<br>mass RIGHT<br>LUNG Left lower lobe<br>nodule LEFT<br>SUPRARENAL GLAND<br>Right adrenal nodule<br>RIGHT | No |
| UK2118 | LUNG Right upper lobe RIGHT | LUNG T1 Right upper lobe RIGHT | Yes |
| | LUNG Right upper lobe RIGHT | LUNG T2 Right upper lobe RIGHT | |
| UK2202 | LUNG Right upper lobe nodule RIGHT | LUNG Right upper lobe nodule RIGHT | Yes |
| UK2206 | LUNG Left lingular metastasis LEFT | LUNG Left lingular<br>metastasis LEFT | Yes |
| | LUNG Lower lobe metastasis LEFT | LUNG lower lobe<br>metastasis LEFT | |
| UK2207 | LUNG Right upper lobe pulmonary mass RIGHT | LUNG Upper lobe pulmonary mass RIGHT | Yes |
| UK2209 | LUNG Right upper lobe lesion RIGHT | LUNG Right upper lobe lesion RIGHT | Yes |
| UK2210 | LYMPH NODE Station 2R right paratracheal node RIGHT | LYMPH NODE Station<br>2R right paratracheal<br>node RIGHT | Yes |
| TITZAGA | LYMPH NODE Right hilar nodal mass RIGHT | LYMPH NODE Right<br>hilar nodal mass RIGHT | 77 |
| UK2211 | LUNG Right upper lobe nodule RIGHT | LUNG Right upper lobe nodule RIGHT | Yes |




| Pt ID | Confirmatory Pre-baseline target lesions (reference scan) | Baseline target lesions | Comments |
|---|---|---|---|
| UK2212 | LYMPH NODE Right Paratracheal<br>Lymph Node RIGHT | LYMPH NODE Right<br>Paratracheal Lymph<br>Node RIGHT | Yes |
| | LYMPH NODE Left Para-aortic Lymph<br>Node LEFT | LYMPH NODE Left<br>Para-aortic Lymph<br>Node LEFT | |
| UK2301 | LUNG Lower lobe LEFT | LUNG Lower lobe<br>LEFT | Yes |
| US3105 | LUNG Left infrahiliar nodule LEFT | LYMPH NODE pre carinal lymph node | No |
| US3108 | BONE Sacrum LEFT | BONE Sacrum LEFT | Yes |
| | LUNG Right posterior apical lesion<br>RIGHT | LUNG Right posterior apical lesion RIGHT | |
| | LUNG Left posterior apical lesion LEFT | LUNG Left posterior<br>apical lesion LEFT | |
| | | BONE Right iliac mass<br>RIGHT | |
| US3109 | LUNG Posterior right upper lobe lesion<br>RIGHT | LUNG Posterior right<br>upper lobe lesion<br>RIGHT | Yes |
| | LUNG Superior segment right lower lobe RIGHT | LUNG Superior segment right lower lobe RIGHT | |
| US3114 | LUNG Left Upper lobe spiculated mass<br>LEFT | LUNG Anterior segment<br>of the right upper lobe<br>RIGHT | Yes, but only the three lesions in bold |
| | LUNG Anterior segment of the right upper lobe RIGHT | OTHER Pleural based<br>mass posterior midlung<br>RIGHT | |
| | OTHER Right Pleura, posterior midlung RIGHT | OTHER Right lateral pleural mass RIGHT | |
| | OTHER Right lateral pleural mass<br>RIGHT | LUNG Right posterior<br>costophrenic angle<br>RIGHT | |
| | | BONE L1 right vertebral body RIGHT | |
| US3120 | LUNG Right Upper lobe mass RIGHT | LUNG Right Middle Lobe mass RIGHT LUNG Right lower lobe | No |
| US3123 | LUNG left upper lobe nodule LEFT | mass RIGHT LUNG left anterior apex spiculated nodule LEFT LUNG left lower lobe | No |
| US3123 | LUNG left upper lobe nodule LEFT | LUNG left anterior apex spiculated nodule LEFT LUNG left lower lobe nodular opacity LEFT LYMPH NODE mediastinal lymph node LIVER right lobe liver RIGHT LIVER second right lobe | No |
| US3123<br>US3401 | LYMPH NODE anterior mediastinal | LUNG left anterior apex spiculated nodule LEFT LUNG left lower lobe nodular opacity LEFT LYMPH NODE mediastinal lymph node LIVER right lobe liver RIGHT | No Yes but only |




| Pt ID | Confirmatory Pre-baseline target lesions (reference scan) | Baseline target lesions | Comments |
|---|---|---|---|
| | | LYMPH NODE anterior | anterior mediastinal |
| | | mediastinal RIGHT | RIGHT |
| | | SUPRARENAL GLAND | |
| | | RIGHT ADRENAL | |
| | | RIGHT | |
| US3402 | LUNG Left Mass LEFT | LUNG Left Mass LEFT | Yes |
| | LUNG Right Mass RIGHT | LUNG Right Mass | |
| | | RIGHT | |




| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

# 5.6.2 Subgroup for Part B (Prior Therapy anti-PD-(L)1-based – cat)

Derivation of previous therapy is provided by Immutep medical team to be integrated in the program based in below categorization.

Previous Therapy = Anti-PD-X + chemo vs Anti-PD-X alone or Anti-PD-X alone + ICI

| Anti-PD-(L)1 | ICI (Immune Checkpoint Inhibitors) | Chemotherapy |
|---|---|---|
| Pembrolizumab | Ipilimumab | Carboplatin |
| Durvalumab | | Cisplatin |
| Nivolumab | | Pemetrexed / Pemetrexed Disodium |
| Atezolizumab | | Gemcitabine |
| Avelumab | | Paclitaxel |


Effective Date: 15th March 2017

Prior Effective Date: 9th October 2016



| Sponsor: | Immutep S.A.S. | Protocol Number: | TACTI-002 (IMP321-<br>P015); Keynote-PN798 |
|---|---|---|---|
|---|---|---|---|

#### 5.7 References

- 1. Simon, R. 1989. Optimal two-stage designs for phase II clinical trials. Control Clin Trials 10(1): 1-10.
- 2. Seymour L, Bogaerts J, Perrone A, et al. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics [published correction appears in Lancet Oncol. 2019 May;20(5):e242]. Lancet Oncol. 2017;18(3):e143-e152. doi:10.1016/S1470-2045(17)30074-8
- 3. Kluger HM, Tawbi HA, Ascierto ML, et al. Defining tumor resistance to PD-1 pathway blockade: recommendations from the first meeting of the SITC Immunotherapy Resistance Taskforce. Journal for ImmunoTherapy of Cancer 2020;8:e000398. doi:10.1136/jitc-2019-000398;Individual patient data analysis to assess modifications to the RECIST criteria. Jan Bogaerts 1, Robert Ford, Dan Sargent, Lawrence H Schwartz, Larry Rubinstein, Denis Lacombe, Elizabeth Eisenhauer, Jaap Verweij, Patrick Therasse, RECIST Working Party. Eur J Cancer. 2009 Jan;45(2):248-60. doi: 10.1016/j.ejca.2008.10.027. Epub 2008 Dec 16.
- 4. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026.
- 5. Saâda-Bouzid, E., et al., Hyperprogression during anti-PD-1/PD-L1 therapy in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Ann Oncol, 2017. 28(7): p. 1605-161;
- 6. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lesley Seymour 1, Jan Bogaerts 2, Andrea Perrone 3, Robert Ford 4, Lawrence H Schwartz 5, Sumithra Mandrekar 6, Nancy U Lin 7, Saskia Litière 2, Janet Dancey 8, Alice Chen 9, F Stephen Hodi 7, Patrick Therasse 10, Otto S Hoekstra 11, Lalitha K Shankar 12, Jedd D Wolchok 13, Marcus Ballinger 14, Caroline Caramella 15, Elisabeth G E de Vries 16, RECIST working group. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2.

Effective Date: 15th March 2017

Prior Effective Date: 9th October 2016

# **Electronic Record and Signature Disclosure**

**DocuSign** 

**Certificate Of Completion** 



**Record Tracking** 

PPD

Signer Events Signature Timestamp

PPD

Signature Adoption: Pre-selected Style Signature ID:

**PPD** 

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure:

Accented: 1/31/2024 2:32:46 PM

**PPD** 

Signer Events Signature Timestamp



**Electronic Record and Signature Disclosure:** 

Accepted: 2/1/2024 4:52:46 AM

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |

**Certified Delivery Events** 



VIEWED

PPD

Status

Timestamp

Sent: 2/1/2024 4:53:21 AM Viewed: 2/1/2024 4:54:54 AM

**Electronic Record and Signature Disclosure:** 

Accented: 2/1/2024 4:54:54 AM

PPD

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent<br>Certified Delivered | Hashed/Encrypted<br>Security Checked | 1/31/2024 9:59:09 AM<br>2/1/2024 4:54:54 AM |
| Signing Complete<br>Completed | Security Checked Security Checked | 2/1/2024 4:53:17 AM<br>2/1/2024 4:54:54 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Fortrea Enterprise (Part 11) (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

# Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### **How to contact Fortrea Enterprise (Part 11):**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

## To advise Fortrea Enterprise (Part 11) of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from Fortrea Enterprise (Part 11)

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Fortrea Enterprise (Part 11)

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to ppD and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Fortrea Enterprise (Part 11) as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Fortrea Enterprise (Part 11) during the course of your relationship with Fortrea Enterprise (Part 11).